CLINICAL TRIAL: NCT03154086
Title: A Phase I, First Time in Human, Two Part, Randomized, Placebo-Controlled, Double-Blind (Sponsor Unblind), Single and Repeat Dose Escalating Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK3352589, a REarranged During Transfection (RET) Growth Factor Receptor Tyrosine Kinase Inhibitor, in Normal Healthy Volunteers
Brief Title: A Phase 1, First Time in Human (FTIH) Study to Evaluate GSK3352589, a REarranged During Transfection (RET) Growth Factor Receptor Tyrosine Kinase Inhibitor, in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 207440
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: REarranged during Transfection
MeSH Terms: conditions — Irritable Bowel Syndrome; Multiple Endocrine Neoplasia Type 2a | interventions — GSK3352589

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg (Experimental): Subjects will receive single oral dose of placebo tablet in Period 1 followed by GSK3352589 5 milligrams (mg) tablet in Period 2 followed by GSK3352589 15 mg tablet in Period 3 followed by GSK3352589 50 mg tablet in Period 4 of Cohort 1 in Part A of the study. Subjects will return for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
  Interventions: Drug: GSK3352589; Drug: Matching Placebo
- Part A:Cohort 1:GSK3352589 2mg/ Placebo/GSK3352589 15mg/50mg (Experimental): Subjects will receive single oral dose of GSK3352589 2 mg tablet in Period 1 followed by Placebo tablet in Period 2 followed by GSK3352589 15 mg tablet in Period 3 followed by GSK3352589 50 mg tablet in Period 4 of Cohort 1 in Part A of the study. Subjects will return for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
  Interventions: Drug: GSK3352589; Drug: Matching Placebo
- Part A:Cohort 1: GSK3352589 2mg/5mg/Placebo/GSK3352589 50mg (Experimental): Subjects will receive single oral dose of GSK3352589 2 mg tablet in Period 1 followed by GSK3352589 5 mg tablet in Period 2 followed by Placebo tablet in Period 3 followed by GSK3352589 50 mg tablet in Period 4 of Cohort 1 in Part A of the study. Subjects will return for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
  Interventions: Drug: GSK3352589; Drug: Matching Placebo
- Part A:Cohort 1: GSK3352589 2mg/5mg/15mg/Placebo (Experimental): Subjects will receive single oral dose of GSK3352589 2 mg tablet in Period 1 followed by GSK3352589 5 mg tablet in Period 2 followed by GSK3352589 15 mg tablet in Period 3 followed by Placebo tablet in Period 4 of Cohort 1 in Part A of the study. Subjects will return for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
  Interventions: Drug: GSK3352589; Drug: Matching Placebo
- Part A:Cohort 2: GSK3352589 25mg Fasted/GSK3352589 25mg Fed (Experimental): Subjects will receive single oral dose of GSK3352589 25 mg tablet in Period 1 (fasted state) and Period 2 (fed state). Subjects will return for their next scheduled dosing Period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
  Interventions: Drug: GSK3352589
- Part A: Cohort 2: Placebo Fasted/Placebo Fed (Experimental): Subjects will receive single oral dose of placebo tablet matching GSK3352589 25 mg in Period 1 (fasted state) and Period 2 (fed state). Subjects will return for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
  Interventions: Drug: Matching Placebo
- Part A:Cohort 3: GSK3352589 150 mg/Placebo (Experimental): Subjects will receive single oral dose of GSK3352589 150 mg tablet in Period 1 followed by placebo tablet matching GSK3352589 150 mg in Period 2 in Cohort 3 of Part A. Subjects will return for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
  Interventions: Drug: GSK3352589; Drug: Matching Placebo
- Part A:Cohort 3: Placebo/GSK3352589 400 mg (Experimental): Subjects will receive single oral dose of placebo tablet matching GSK3352589 400 mg in Period 1 followed by single oral dose of GSK3352589 400 mg tablet in Period 2 in Cohort 3 of Part A. Subjects will return for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
  Interventions: Drug: GSK3352589; Drug: Matching Placebo
- Part A:Cohort 3: GSK3352589 150mg/GSK3352589 400mg (Experimental): Subjects will receive single oral dose of GSK3352589 150 mg tablet in Period 1 followed by GSK3352589 400 mg tablet in Period 2 in Cohort 3 of Part A. Subjects will return for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
  Interventions: Drug: GSK3352589
- Part B: GSK3352589 (Experimental): Subjects will receive repeat oral doses of GSK3352589 of 5 mg, 15 mg, 50 mg, 100 mg or 200 mg twice daily administered for 14 days.
  Interventions: Drug: GSK3352589
- Part B: Placebo (Placebo Comparator): Subjects will receive repeat oral doses of placebo twice a day tablet administered for 14 days.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: GSK3352589 — It will be available in the dose of 1, 5, 25 and 100 mg tablet for oral administration.
  Arms: Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg; Part A:Cohort 1: GSK3352589 2mg/5mg/15mg/Placebo; Part A:Cohort 1: GSK3352589 2mg/5mg/Placebo/GSK3352589 50mg; Part A:Cohort 1:GSK3352589 2mg/ Placebo/GSK3352589 15mg/50mg; Part A:Cohort 2: GSK3352589 25mg Fasted/GSK3352589 25mg Fed; Part A:Cohort 3: GSK3352589 150 mg/Placebo; Part A:Cohort 3: GSK3352589 150mg/GSK3352589 400mg; Part A:Cohort 3: Placebo/GSK3352589 400 mg; Part B: GSK3352589
Drug: Matching Placebo — It will be available across all strengths to match active drug in the form of tablet for oral administration.
  Arms: Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg; Part A: Cohort 2: Placebo Fasted/Placebo Fed; Part A:Cohort 1: GSK3352589 2mg/5mg/15mg/Placebo; Part A:Cohort 1: GSK3352589 2mg/5mg/Placebo/GSK3352589 50mg; Part A:Cohort 1:GSK3352589 2mg/ Placebo/GSK3352589 15mg/50mg; Part A:Cohort 3: GSK3352589 150 mg/Placebo; Part A:Cohort 3: Placebo/GSK3352589 400 mg; Part B: Placebo

SUMMARY:
This FTIH study is designed to assess the safety, tolerability and pharmacokinetic (PK) of escalating single and repeat oral doses of GSK3352589 in normal healthy volunteers. This is a randomized, double-blind (sponsor unblinded), placebo controlled, dose escalation study that will have two parts; Part A and Part B.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. - History of regular bowel habits
* Male or Female of non-childbearing potential.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions.

Exclusion Criteria:

* ALT and bilirubin >1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Previous Diagnosis of IBS
* Estimated Glomerular Filtration Rate <60 millilter per minute per 1.73 square meter (mL/min/1.73m^2)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* History of Gastroesophageal reflux disease (GERD), dyspepsia, Gastrointestinal (GI) bleeding, diverticulitis, diverticular stricture or other intestinal strictures, GI surgery that could affect motility
* Unwillingness or inability to follow the procedures outlined in the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reedy BA, O'Connor-Semmes R, Hacquoil K, Gorycki P, Verticelli A, Molga A. First-in-Human Study for a Selective Rearranged During Transfection Tyrosine Kinase Inhibitor, GSK3352589, to Investigate the Safety, Tolerability, and Pharmacokinetics in Healthy Volunteers. Clin Pharmacol Drug Dev. 2021 Apr;10(4):334-345. doi: 10.1002/cpdd.911. Epub 2021 Feb 19. PMID 33606922

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two-part study. Part A was a single dose escalating and Part B was a repeat dose escalating. Participants participated in either Part A or Part B of the study. This was a single center study, conducted at one site in Australia.
Pre-assignment Details: A total number of 28 participants were enrolled in Part A and 40 participants were enrolled in Part B of the study. Participants in Part A, participated in one of the 3 Cohorts in Part A and Part B participants participated in one of the 5 Cohorts in Part B.
Groups:
- Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg: Participants received single oral dose of placebo tablet in Period 1 followed by GSK3352589 5 milligrams (mg) tablet in Period 2 followed by GSK3352589 15 mg tablet in Period 3 followed by GSK3352589 50 mg tablet in Period 4 of Cohort 1 in Part A of the study. Participants returned for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
- Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg: Participants received single oral dose of GSK3352589 2 mg tablet in Period 1 followed by Placebo tablet in Period 2 followed by GSK3352589 15 mg tablet in Period 3 followed by GSK3352589 50 mg tablet in Period 4 of Cohort 1 in Part A of the study. Participants returned for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
- Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg: Participants received single oral dose of GSK3352589 2 mg tablet in Period 1 followed by GSK3352589 5 mg tablet in Period 2 followed by Placebo tablet in Period 3 followed by GSK3352589 50 mg tablet in Period 4 of Cohort 1 in Part A of the study. Participants returned for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
- Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo: Participants received single oral dose of GSK3352589 2 mg tablet in Period 1 followed by GSK3352589 5 mg tablet in Period 2 followed by GSK3352589 15 mg tablet in Period 3 followed by Placebo tablet in Period 4 of Cohort 1 in Part A of the study. Participants returned for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
- Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed: Participants received single oral dose of GSK3352589 25 mg tablet in Period 1 (fasted state) and in Period 2 (fed state). Participants returned for their next scheduled dosing Period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
- Part A: Cohort 2: Placebo Fasted/Placebo Fed: Participants received single oral dose of placebo tablet matching GSK3352589 25 mg in Period 1 (fasted state) and in Period 2 (fed state). Participants returned for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
- Part A:Cohort 3: GSK3352589 150 mg/Placebo: Participants received single oral dose of GSK3352589 150 mg tablet in Period 1 followed by placebo tablet matching GSK3352589 150 mg in Period 2 in Cohort 3 of Part A. Participants returned for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
- Part A:Cohort 3: Placebo /GSK3352589 400 mg: Participants received single oral dose of placebo tablet matching GSK3352589 400 mg in Period 1 followed by single oral dose of GSK3352589 400 mg tablet in Period 2 in Cohort 3 of Part A. Participants returned for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
- Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg: Participants received single oral dose of GSK3352589 150 mg tablet in Period 1 followed by GSK3352589 400 mg tablet in Period 2 in Cohort 3 of Part A. Participants returned for their next scheduled dosing period approximately 14 days (wash out period) after administration of the study drug during the prior dosing period.
- Part B: Placebo BID: Participants received repeat oral doses of placebo BID (twice a day) tablet administered for 14 days in Part B of the study.
- Part B: GSK3352589 5 mg BID: Participants received repeat oral doses of GSK3352589 5 mg BID tablet administered for 14 days in Part B of the study.
- Part B: GSK3352589 15 mg BID: Participants received repeat oral doses of GSK3352589 15 mg BID tablet administered for 14 days in Part B of the study.
- Part B: GSK3352589 50 mg BID: Participants received repeat oral doses of GSK3352589 50 mg BID tablet administered for 14 days in Part B of the study.
- Part B: GSK3352589 100 mg BID: Participants received repeat doses of GSK3352589 100 mg BID administered for 14 days in Part B of the study.
- Part B: GSK3352589 200 mg BID: Participants received repeat doses of GSK3352589 200 mg BID administered for 14 days in Part B of the study.
Period: Part A: Cohort1 Period1 (Up to 3 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort1 Washout1 (Up to 14 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort1 Period2 (Up to 3 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 2 | 2 | 2 | 2 (One replacement participant (par) was enrolled and dosed) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA: Cohort1 Washout2 (Up to 14 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort1 Period3 (Up to 3 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 2 | 2 (One replacement par was enrolled and dosed) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort1 Washout3 (Up to 14 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort1 Period4 (Up to 3 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 3 (1 par was not dosed on day of dosing due to elevated lab; hence 1 replacement was enrolled and dosed) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort2 Period1 (Up to 3 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort2 Washout1 (Up to 14 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort2 Period2 (Up to 3 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort3 Period1 (Up to 3 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort3 Washout1 (Up to 14 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Cohort3 Period2 (Up to 3 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 (1 par was unwell on Day-1 of Period 2 and discontinued; hence,1 replacement was enrolled and dosed) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (Up to 25 Days)
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 6 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 5 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1: Placebo/GSK3352589 5mg/15mg/50mg | Part A:Cohort 1:GSK3352589 2mg/Placebo/GSK3352589 15mg/50mg | Part A:Cohort 1: GSK3352589 2mg/ 5mg/Placebo/ GSK3352589 50mg | Part A:Cohort 1:GSK3352589 2mg/5mg/15mg/Placebo | Part A:Cohort 2:GSK3352589 25 mg Fasted/GSK3352589 25 mg Fed | Part A: Cohort 2: Placebo Fasted/Placebo Fed | Part A:Cohort 3: GSK3352589 150 mg/Placebo | Part A:Cohort 3: Placebo /GSK3352589 400 mg | Part A:Cohort 3: GSK3352589 150 mg/GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID | Total
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 6 | 2 | 2 | 2 | 5 | 10 | 6 | 6 | 6 | 6 | 6 | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (14.00) | 26.7 (4.73) | 33.5 (9.19) | 41.0 (5.20) | 29.7 (8.57) | 34.5 (3.54) | 40.5 (7.78) | 44.5 (0.71) | 28.8 (7.43) | 25.5 (5.40) | 30.8 (8.11) | 33.3 (8.45) | 23.3 (2.88) | 23.7 (4.59) | 32.2 (11.20) | 30.5 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Male | 3 | 3 | 1 | 3 | 6 | 2 | 2 | 2 | 5 | 10 | 6 | 6 | 6 | 6 | 5 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Native-Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 10
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 3 | 3 | 1 | 2 | 6 | 2 | 2 | 1 | 3 | 8 | 5 | 5 | 4 | 5 | 5 | 55
  Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Serious Adverse Events (SAEs) and Non-SAEs in Cohort 1
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or other situations as per medical or scientific judgment.
Time Frame: Up to 64 days in Cohort 1
Population: Safety Population comprised of all randomized participants who received at least one dose of study medication and was based on the actual treatment received, if this differed from that to which the participant was randomized.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Cohort 1: Placebo: Participants received placebo tablet matching GSK3352589 orally in one of the Periods of Cohort 1 in Part A of the study.
- Part A: Cohort 1: GSK3352589 2 mg: Participants received GSK3352589 2 mg tablet orally in Period 1 of Cohort 1 in Part A of the study.
- Part A: Cohort 1: GSK3352589 5 mg: Participants received GSK3352589 5 mg tablet orally in Period 2 of Cohort 1 in Part A of the study.
- Part A: Cohort 1: GSK3352589 15 mg: Participants received GSK3352589 15 mg tablet orally in Period 3 of Cohort 1 in Part A of the study.
- Part A: Cohort 1: GSK3352589 50 mg: Participants received GSK3352589 50 mg tablet in Period 4 of Cohort 1 in Part A of the study.
Arm/Group | Part A: Cohort 1: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 5
Participants
  Any SAE | 0 | 1 | 0 | 0 | 0
  Any non-SAE | 3 | 5 | 3 | 2 | 2

2. Primary Outcome: Part A: Number of Participants With SAEs and Non-SAEs in Cohort 2
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or other situations as per medical or scientific judgment.
Time Frame: Up to 30 days in Cohort 2
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Cohort 2: Fasted Placebo: Participants received placebo tablet matching GSK3352589 without food in Period 1 of Cohort 2 in Part A of the study.
- Part A: Cohort 2: Fed Placebo: Participants received placebo tablet matching GSK3352589 with food in Period 2 of Cohort 2 in Part A of the study.
- Part A: Cohort 2: GSK3352589 Fasted 25 mg: Participants received GSK3352589 25 mg tablet without food in Period 1 of Cohort 1 in Part A of the study.
- Part A: Cohort 2: GSK3352589 Fed 25 mg: Participants received GSK3352589 25 mg tablet with food in Period 2 of Cohort 1 in Part A of the study.
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Participants
  Any SAE | 0 | 0 | 0 | 0
  Any non-SAE | 1 | 0 | 3 | 1

3. Primary Outcome: Part A: Number of Participants With SAEs and Non-SAEs in Cohort 3
Description: as for outcome 2
Time Frame: Up to 30 days in Cohort 3
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Cohort 3: Placebo: Participants received placebo tablet matching GSK3352589 in one of the Periods of Cohort 3 in Part A of the study.
- Part A: Cohort 3: GSK3352589 150 mg: Participants received GSK3352589 150 mg tablet in Period 1 of Cohort 3 in Part A of the study.
- Part A: Cohort 3: GSK3352589 400 mg: Participants received GSK3352589 400 mg tablet in Period 2 of Cohort 3 in Part A of the study.
Arm/Group | Part A: Cohort 3: Placebo | Part A: Cohort 3: GSK3352589 150 mg | Part A: Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 4 | 6 | 5
Participants
  Any SAE | 0 | 0 | 0
  Any non-SAE | 2 | 3 | 1

4. Primary Outcome: Part B: Number of Participants With SAEs and Non-SAEs
Description: as for outcome 2
Time Frame: Up to 25 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Placebo BID: Participants received repeat doses of placebo BID administered for 14 days in Part B of the study.
- Part B: GSK3352589 5 mg BID: Participants received repeat doses of GSK3352589 5 mg BID administered for 14 days in Part B of the study.
- Part B: GSK3352589 15 mg BID: Participants received repeat doses of GSK3352589 15 mg BID administered for 14 days in Part B of the study.
- Part B: GSK3352589 50 mg BID: Participants received repeat doses of GSK3352589 50 mg BID administered for 14 days in Part B of the study.
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0
  Any non-SAE | 9 | 5 | 6 | 2 | 5 | 5

5. Primary Outcome: Part A: Number of Participants With Abnormal Findings After Physical Examination in Cohort 1
Description: A complete physical examination will include, at a minimum, assessments of the skin, cardiovascular, respiratory, gastrointestinal and neurological systems. Brief symptom directed physical examination included, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). Number of participants with clinically significant abnormal physical examination findings have been presented.
Time Frame: Up to 64 days in Cohort 1
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part A: Number of Participants With Abnormal Findings After Physical Examination in Cohort 2
Description: A complete physical examination included, at a minimum, assessments of the skin, cardiovascular, respiratory, gastrointestinal and neurological systems. Brief symptom directed physical examination included, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). Number of participants with clinically significant abnormal physical examination findings have been presented.
Time Frame: Up to 30 days in Cohort 2
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Participants | 0 | 0 | 0 | 0

7. Primary Outcome: Part A: Number of Participants With Abnormal Findings After Physical Examination in Cohort 3
Description: as for outcome 6
Time Frame: Up to 30 days in Cohort 3
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 3: Placebo | Part A: Cohort 3: GSK3352589 150 mg | Part A: Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 4 | 6 | 5
Participants | 0 | 0 | 1

8. Primary Outcome: Part B: Number of Participants With Abnormal Findings After Physical Examination
Description: as for outcome 6
Time Frame: Up to 25 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Part A: Number of Participants With Abnormal Electrocardiogram (ECG) Findings in Cohort 1 and Cohort 3
Description: Triplicate 12-lead ECGs were obtained at indicated time points during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT corrected (QTc) intervals. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Baseline is defined as the last available, non-missing mean value of triplicate assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). The number of participants with abnormal clinically significant (CS) and not clinically significant (NCS) findings for ECG parameters have been presented.
Time Frame: Baseline (Pre-dose on Day 1), Day 1 (1, 4, 12 Hours Post-dose), Day 2
Population: Safety population. In Cohort 1 and 3, participants were dosed in similar single ascending doses, cross-over sequences. Hence, combined totals for placebo arm is presented as pre-specified in protocol and reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Cohort 1 and 3: Placebo: Participants received placebo tablet matching GSK3352589 in one of the Periods of Cohort 1 and Cohort 3 in Part A of the study.
- Part A:Cohort 3: GSK3352589 150 mg: Participants received GSK3352589 150 mg tablet in Period 1 of Cohort 3 in Part A of the study.
- Part A:Cohort 3: GSK3352589 400 mg: Participants received GSK3352589 400 mg tablet in Period 2 of Cohort 3 in Part A of the study.
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Participants
  Baseline (Day 1; Pre-dose); Abnormal NCS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline (Day 1; Pre-dose); Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1; 1 Hour Post-dose; Abnormal NCS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1; 1 Hour Post-dose; Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1; 4 Hours Post-dose; Abnormal NCS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1; 4 Hours Post-dose; Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1; 12 Hours Post-dose; Abnormal NCS | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Day 1; 12 Hours Post-dose; Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 2; Abnormal NCS | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Day 2; Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Part A: Number of Participants With Abnormal ECG Findings in Cohort 2
Description: Triplicate 12-lead ECGs were obtained at indicated time points during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Baseline is defined as the last available, non-missing mean value of triplicate assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). The number of participants with abnormal CS and NCS findings for ECG parameters have been presented.
Time Frame: Baseline (Pre-dose on Day 1), Day 1 (1, 4, 12 Hours Post-dose), Day 2
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Participants
  Baseline (Day 1; Pre-dose); Abnormal NCS | 0 | 0 | 0 | 0
  Baseline; (Day 1;pre dose); Abnormal CS | 0 | 0 | 0 | 0
  Day 1; 1 Hour Post-dose; Abnormal NCS | 0 | 0 | 0 | 0
  Day 1; 1 Hour Post-dose; Abnormal CS | 0 | 0 | 0 | 0
  Day 1; 4 Hours Post-dose; Abnormal NCS | 0 | 0 | 0 | 0
  Day 1; 4 Hours Post-dose; Abnormal CS | 0 | 0 | 0 | 0
  Day 1; 12 Hours Post-dose; Abnormal NCS | 0 | 0 | 0 | 0
  Day 1; 12 Hours Post-dose; Abnormal CS | 0 | 0 | 0 | 0
  Day 2; Abnormal NCS | 0 | 0 | 0 | 0
  Day 2; Abnormal CS | 0 | 0 | 0 | 0

11. Primary Outcome: Part B: Number of Participants With Abnormal ECG Findings
Description: Triplicate 12-lead ECGs were obtained at indicated time points during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Baseline is defined as the last available, non-missing mean value of triplicate assessment prior to the first administration of study drug. The number of participants with abnormal CS and NCS findings for ECG parameters have been presented.
Time Frame: Baseline (Pre-dose on Day 1), Day 1 (4 Hours Post-dose), Day 7 (Pre-dose, 4 Hours Post-dose), Day 14 (Pre-dose, 4 Hours Post-dose), Follow-up (Day 25)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants
  Baseline (Day 1; Pre-dose); Abnormal NCS | 0 | 0 | 0 | 0 | 0 | 0
  Baseline (Day 1; Pre-dose); Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0
  Day 1; 4 Hours Post-dose; Abnormal NCS | 0 | 0 | 0 | 0 | 0 | 1
  Day 1; 4 Hours Post-dose; Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0
  Day 7; Pre-dose; Abnormal NCS | 0 | 0 | 0 | 0 | 1 | 0
  Day 7; Pre-dose; Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0
  Day 7; 4 Hours Post-dose; Abnormal NCS | 0 | 0 | 0 | 0 | 0 | 0
  Day 7; 4 Hours Post-dose; Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0
  Day 14; Pre-dose; Abnormal NCS | 0 | 0 | 0 | 0 | 0 | 0
  Day 14; Pre-dose; Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0
  Day 14; 4 Hours Post-dose; Abnormal NCS | 1 | 0 | 0 | 0 | 0 | 0
  Day 14; 4 Hours Post-dose; Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0
  Follow-up (Day 25); Abnormal NCS | 1 | 0 | 1 | 0 | 0 | 0
  Follow-up (Day 25); Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Part A: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in Cohort 1 and Cohort 3
Description: Blood pressure of participants was measured at indicated time points in a supine position after 5 minutes rest. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Pre-dose on Day 1), Day 1 (1, 4, 12 Hours Post-dose), Day 2 and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Millimeters of mercury
  SBP; Day 1; 1 Hour Post dose | -1.25 (9.61) | -1.75 (4.71) | -2.08 (11.72) | 3.00 (9.72) | -2.70 (12.26) | 1.58 (5.55) | -0.10 (3.45)
  SBP; Day 1; 4 Hours Post dose | -1.29 (11.32) | -5.83 (5.86) | -1.33 (13.56) | 3.75 (11.04) | -3.60 (14.72) | -1.75 (3.27) | 1.40 (1.29)
  SBP; Day 1; 12 Hours Post dose | 2.21 (8.65) | -3.83 (10.11) | 1.08 (11.33) | 3.00 (10.39) | 3.10 (9.15) | 1.33 (4.07) | 3.90 (6.69)
  SBP; Day 2 | -2.42 (10.00) | -4.50 (5.74) | -1.42 (9.77) | -2.17 (10.87) | -3.40 (7.54) | 1.50 (2.53) | -5.00 (5.78)
  SBP; Day 3 | -3.63 (11.05) | -8.67 (5.12) | -0.42 (16.59) | 1.92 (7.05) | -3.30 (10.12) | 0.67 (4.17) | 0.60 (5.90)
  DBP; Day 1; 1 Hour Post dose | -0.54 (5.62) | -0.67 (3.89) | 1.75 (4.71) | 1.08 (7.34) | 1.00 (10.31) | 0.33 (4.01) | 4.20 (2.59)
  DBP; Day 1; 4 Hours Post dose | 2.04 (5.87) | -0.42 (5.33) | -1.83 (5.39) | 2.25 (9.95) | -2.10 (6.07) | 1.17 (4.77) | 6.50 (2.06)
  DBP; Day 1; 12 Hours Post dose | -2.92 (5.67) | -4.42 (6.58) | -3.08 (5.29) | -5.75 (5.33) | -4.10 (8.13) | -1.08 (5.30) | 0.40 (7.99)
  DBP; Day 2 | -2.13 (4.71) | -2.58 (7.91) | -2.25 (4.10) | -1.17 (4.01) | -5.40 (3.44) | -0.17 (5.34) | 3.60 (4.92)
  DBP; Day 3 | 1.13 (6.30) | -2.67 (7.72) | 2.67 (5.65) | -1.50 (6.43) | -2.20 (4.27) | 0.75 (4.97) | 3.80 (4.91)

13. Primary Outcome: Part A: Change From Baseline in SBP and DBP in Cohort 2
Description: as for outcome 12
Time Frame: Baseline (Pre-dose on Day 1), Day 1 (1, 4, 12 Hours Post-dose), Day 2 and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Millimeters of mercury
  SBP; Day 1; 1 Hour Post dose | 3.75 (3.89) | 6.00 (8.49) | 3.75 (9.68) | -6.58 (9.91)
  SBP; Day 1; 4 Hours Post dose | -1.75 (1.06) | -6.50 (9.19) | -5.17 (11.44) | -6.25 (10.30)
  SBP; Day 1; 12 Hours Post dose | 1.75 (9.55) | 10.75 (15.91) | 1.50 (10.84) | 1.50 (11.66)
  SBP; Day 2 | -6.75 (5.30) | -3.75 (4.60) | -7.58 (5.18) | -5.00 (9.77)
  SBP; Day 3 | -0.25 (0.35) | 6.75 (10.96) | -4.50 (8.06) | 1.00 (7.54)
  DBP; Day 1; 1 Hour Post dose | 1.25 (3.89) | -5.75 (2.47) | 1.67 (6.23) | -4.25 (5.67)
  DBP; Day 1; 4 Hours Post dose | -3.25 (3.18) | -5.00 (3.54) | -1.67 (7.10) | -4.75 (5.99)
  DBP; Day 1; 12 Hours Post dose | -5.25 (2.47) | -3.00 (2.83) | -2.67 (6.92) | -6.00 (6.87)
  DBP; Day 2 | -3.50 (2.12) | -5.25 (6.72) | -1.92 (4.41) | -2.75 (3.49)
  DBP; Day 3 | 1.50 (8.49) | 0.75 (7.42) | 3.58 (6.94) | 2.08 (5.01)

14. Primary Outcome: Part B: Change From Baseline in SBP and DBP
Description: Blood pressure of participants was measured at indicated time points in a supine position after 5 minutes rest. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Pre-dose on Day 1), Day 1 (4 Hours Post-dose), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7 (Pre-dose, 4 Hours Post-dose), Day 8, Day 9, Day 10, Day 11, Day 12, Day 13, Day 14 (Pre-dose, 4 Hours Post-dose), Day 15, Follow-up (Day 25)
Population: Safety population. Only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Millimeters of mercury
  SBP; Day 1; 4 Hours Post dose; n=10,6,6,6,6,6 | -4.70 (7.00) | -1.83 (6.59) | -2.33 (6.01) | 1.17 (10.69) | -2.33 (11.79) | -8.08 (7.39)
  SBP; Day 2; n=10,6,6,6,6,6 | -7.35 (5.61) | -6.25 (5.37) | -5.75 (7.37) | -2.33 (13.01) | -4.08 (12.69) | -9.42 (11.58)
  SBP; Day 3; n=10,6,6,6,6,6 | -5.90 (6.50) | -5.25 (13.97) | -1.42 (6.42) | -9.83 (18.11) | -6.83 (11.57) | -5.58 (5.24)
  SBP; Day 4; n=10,6,6,6,6,6 | -7.75 (6.91) | -5.83 (9.23) | 0.83 (8.88) | -0.08 (15.46) | -9.08 (11.13) | -9.42 (6.26)
  SBP; Day 5; n=10,6,6,6,6,6 | -8.55 (8.39) | -7.00 (5.85) | -1.08 (5.39) | -9.33 (18.90) | -3.92 (14.39) | -11.17 (8.52)
  SBP; Day 6; n=10,6,6,6,6,6 | -9.65 (6.93) | -5.33 (8.52) | -5.42 (4.25) | -6.50 (13.10) | -4.08 (16.53) | -10.33 (15.03)
  SBP; Day 7, Pre-dose; n=10,6,6,6,6,6 | -7.25 (8.36) | -9.75 (6.57) | -7.83 (5.85) | -7.83 (14.75) | -3.50 (10.48) | -3.92 (13.91)
  SBP; Day 7, 4 Hours Post-dose; n=10,6,6,6,6,6 | -9.00 (5.61) | -6.92 (6.50) | -6.67 (7.93) | -6.92 (10.58) | -5.92 (15.81) | -7.50 (14.55)
  SBP; Day 8; n=10,6,6,6,6,6 | -8.95 (5.71) | -6.00 (9.87) | -7.67 (14.50) | -4.50 (10.31) | -8.00 (9.98) | -4.75 (10.01)
  SBP; Day 9; n=10,6,6,6,6,6 | -11.90 (9.74) | 0.67 (11.89) | -5.83 (5.19) | -11.08 (15.23) | -8.33 (11.99) | -9.00 (13.70)
  SBP; Day 10; n=10,6,6,6,6,6 | -7.15 (7.34) | -5.67 (7.15) | -1.67 (6.25) | -7.67 (15.08) | -9.50 (13.57) | -15.67 (18.97)
  SBP; Day 11; n=10,6,6,6,6,6 | -8.60 (8.03) | -5.00 (9.42) | -3.83 (14.31) | -7.25 (16.23) | -8.42 (10.95) | -9.50 (10.31)
  SBP; Day 12; n=10,6,6,6,6,6 | -8.50 (9.06) | -5.58 (10.74) | -0.08 (10.03) | -4.00 (18.10) | -9.33 (13.52) | -4.25 (12.50)
  SBP; Day 13; n=10,6,6,6,6,6 | -9.15 (7.63) | -5.33 (10.30) | -1.58 (6.96) | -6.67 (17.26) | -8.08 (16.69) | -6.58 (9.84)
  SBP; Day 14, Pre-dose; n=10,6,6,6,6,6 | -6.90 (9.73) | -5.42 (7.64) | -0.25 (3.76) | -1.83 (15.28) | 0.83 (10.93) | -9.50 (6.98)
  SBP; Day 14, 4 Hours Post-dose; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  SBP; Day 14, 4 Hours Post-dose; n=10,5,6,6,6,6 | -5.15 (9.48) | -8.50 (8.12) | 0.50 (7.13) | -13.00 (13.90) | -0.25 (13.15) | -5.67 (8.64)
  SBP; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  SBP; Day 15; n=10,5,6,6,6,6 | -6.05 (10.20) | -1.00 (6.78) | 8.08 (8.11) | -5.92 (14.17) | 2.67 (13.53) | -5.42 (8.46)
  SBP; Follow-up (Day 25); n=10,6,6,6,6,6 | -6.85 (9.32) | -4.42 (11.63) | -3.67 (7.74) | 0.08 (11.00) | -1.08 (12.64) | -2.83 (7.81)
  DBP; Day 1; 4 Hours Post dose; n=10,6,6,6,6,6 | -4.90 (5.78) | -2.17 (5.27) | -1.42 (6.92) | -2.08 (5.56) | -5.00 (7.06) | -3.33 (6.77)
  DBP; Day 2; n=10,6,6,6,6,6 | -6.05 (4.83) | 1.50 (9.84) | -1.67 (5.60) | -3.67 (8.22) | -3.17 (7.47) | -2.25 (8.85)
  DBP; Day 3; n=10,6,6,6,6,6 | -3.30 (5.30) | 0.08 (6.64) | -2.75 (4.91) | -3.50 (6.19) | -5.00 (6.54) | -2.17 (7.16)
  DBP; Day 4; n=10,6,6,6,6,6 | -7.05 (6.89) | -0.58 (10.28) | -1.33 (4.54) | -3.00 (5.93) | -3.33 (2.82) | -3.67 (6.68)
  DBP; Day 5; n=10,6,6,6,6,6 | -7.80 (9.26) | -1.67 (5.67) | -4.17 (3.92) | -8.25 (7.90) | -3.58 (6.44) | -3.33 (9.36)
  DBP; Day 6; n=10,6,6,6,6,6 | -10.20 (7.37) | -1.67 (4.83) | -3.25 (6.02) | -7.25 (5.82) | -3.00 (7.54) | -6.67 (7.94)
  DBP; Day 7, Pre-dose; n=10,6,6,6,6,6 | -7.20 (7.52) | -4.17 (4.67) | -6.75 (7.76) | -5.17 (5.83) | 4.58 (3.99) | 0.33 (8.68)
  DBP; Day 7, 4 Hours Post-dose; n=10,6,6,6,6,6 | -8.65 (7.04) | -3.75 (4.12) | -5.92 (4.62) | -6.83 (6.12) | -2.75 (7.06) | -3.67 (10.24)
  DBP; Day 8; n=10,6,6,6,6,6 | -8.20 (6.86) | -1.75 (9.42) | -5.50 (9.49) | -2.75 (8.93) | -1.25 (4.47) | -4.42 (7.49)
  DBP; Day 9; n=10,6,6,6,6,6 | -10.00 (8.36) | -1.08 (8.67) | -3.08 (4.19) | -8.00 (9.17) | -6.75 (7.13) | -4.42 (6.73)
  DBP; Day 10; n=10,6,6,6,6,6 | -5.35 (8.93) | 1.50 (4.71) | -3.00 (7.22) | -5.25 (6.26) | -2.42 (8.75) | -6.50 (12.08)
  DBP; Day 11; n=10,6,6,6,6,6 | -6.80 (10.14) | -1.25 (8.60) | -4.58 (7.37) | -6.25 (7.01) | -5.08 (4.73) | -3.92 (7.21)
  DBP; Day 12; n=10,6,6,6,6,6 | -6.95 (5.44) | -2.67 (8.65) | -1.42 (4.44) | -5.42 (7.81) | -2.00 (3.79) | -0.50 (7.62)
  DBP; Day 13; n=10,6,6,6,6,6 | -7.55 (8.26) | -1.42 (10.70) | -2.50 (5.13) | -2.92 (8.23) | -1.08 (5.70) | -2.67 (8.17)
  DBP; Day 14, Pre-dose; n=10,6,6,6,6,6 | -6.10 (7.05) | -4.25 (6.19) | 0.17 (5.69) | -3.58 (5.10) | 2.67 (3.66) | -0.83 (7.77)
  DBP; Day 14, 4 Hours Post-dose; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  DBP; Day 14, 4 Hours Post-dose; n=10,5,6,6,6,6 | -6.65 (7.12) | -6.80 (8.25) | -3.58 (4.87) | -8.83 (7.45) | 5.00 (5.68) | 0.33 (8.85)
  DBP; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  DBP; Day 15; n=10,5,6,6,6,6 | -6.75 (10.22) | 1.30 (7.13) | 2.00 (7.47) | -5.67 (6.47) | 2.00 (8.40) | -4.08 (7.28)
  DBP; Follow-up (Day 25); n=10,6,6,6,6,6 | -5.85 (8.87) | -3.92 (7.56) | -1.75 (5.10) | -1.75 (8.62) | 1.00 (5.06) | -1.17 (10.63)

15. Primary Outcome: Part A: Change From Baseline in Pulse Rate in Cohort 1 and Cohort 3
Description: Pulse rate of participants was measured at indicated time points in a supine position after 5 minutes rest. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Pre-dose on Day 1), Day 1 (1, 4, 12 Hours Post-dose), Day 2 and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Beats per minute
  Day 1; 1 Hour Post dose | -3.79 (6.30) | -3.25 (4.39) | -3.00 (6.66) | -3.25 (6.93) | -4.00 (7.44) | -2.75 (5.69) | -3.20 (5.38)
  Day 1; 4 Hours Post dose | -6.42 (5.91) | -4.92 (5.98) | -4.67 (6.59) | -0.75 (7.96) | -6.90 (5.03) | -3.67 (4.70) | -3.40 (3.17)
  Day 1; 12 Hours Post dose | 2.38 (6.34) | 0.75 (3.40) | 5.83 (6.04) | 6.00 (3.10) | 0.40 (8.93) | 2.33 (3.88) | 2.40 (6.44)
  Day 2 | -1.46 (9.11) | -3.33 (7.77) | -2.42 (6.90) | 2.08 (4.57) | -3.60 (7.21) | -2.83 (2.14) | -1.60 (3.60)
  Day 3 | 0.54 (7.17) | -0.08 (10.84) | -1.75 (9.49) | 0.50 (7.06) | -2.50 (10.62) | -2.08 (5.44) | 0.50 (5.15)

16. Primary Outcome: Part A: Change From Baseline in Pulse Rate in Cohort 2
Description: as for outcome 15
Time Frame: Baseline (Pre-dose on Day 1), Day 1 (1, 4, 12 Hours Post-dose), Day 2 and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Beats per minute
  Day 1; 1 Hour Post dose | 1.50 (1.41) | 7.50 (0.71) | 0.42 (4.98) | 9.08 (4.33)
  Day 1; 4 Hours Post dose | 1.75 (2.47) | -1.00 (2.12) | -1.33 (3.87) | 2.75 (3.95)
  Day 1; 12 Hours Post dose | 7.00 (2.12) | 9.25 (0.35) | 9.33 (3.42) | 7.92 (2.76)
  Day 2 | 1.25 (3.89) | 3.00 (4.24) | 4.33 (4.74) | 3.17 (5.39)
  Day 3 | 8.00 (4.95) | 4.75 (3.18) | 6.92 (7.12) | 7.58 (8.29)

17. Primary Outcome: Part B: Change From Baseline in Pulse Rate
Description: Pulse rate of participants was measured at indicated time points in a supine position after 5 minutes rest. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Beats per minute
  Day 1; 4 Hours Post dose; n=10,6,6,6,6,6 | -1.55 (4.75) | -0.42 (8.65) | -2.25 (4.16) | -3.58 (4.90) | -1.17 (7.13) | -3.42 (5.74)
  Day 2; n=10,6,6,6,6,6 | 3.35 (7.07) | 2.50 (10.80) | -0.25 (5.52) | 0.50 (8.63) | -2.67 (7.28) | 0.08 (6.41)
  Day 3; n=10,6,6,6,6,6 | 4.85 (4.53) | 3.33 (7.05) | 0.58 (5.62) | 1.08 (8.34) | -6.92 (8.45) | -2.25 (5.35)
  Day 4; n=10,6,6,6,6,6 | 3.25 (8.47) | 2.42 (10.53) | -1.67 (3.80) | 1.33 (9.10) | 2.58 (9.16) | -0.17 (6.77)
  Day 5; n=10,6,6,6,6,6 | -0.25 (6.03) | -1.17 (9.03) | 2.75 (6.83) | 1.92 (9.09) | -0.25 (9.96) | 3.92 (10.11)
  Day 6; n=10,6,6,6,6,6 | -0.50 (5.33) | 5.42 (11.74) | -0.33 (8.94) | -1.33 (8.24) | 0.08 (9.04) | -2.67 (8.05)
  Day 7, Pre-dose; n=10,6,6,6,6,6 | -1.55 (5.23) | 0.25 (8.30) | -0.25 (10.24) | -0.75 (5.66) | 0.50 (9.44) | -0.25 (5.40)
  Day 7, 4 Hours Post-dose; n=10,6,6,6,6,6 | 0.20 (4.82) | 3.75 (10.14) | -5.08 (5.38) | -0.58 (5.52) | -1.25 (7.29) | 1.17 (6.63)
  Day 8; n=10,6,6,6,6,6 | 0.55 (7.37) | 1.42 (9.06) | 1.42 (6.15) | 2.08 (7.28) | -0.17 (10.75) | 5.83 (6.93)
  Day 9; n=10,6,6,6,6,6 | 1.05 (8.59) | 2.58 (7.01) | 0.83 (5.91) | 2.50 (5.59) | -4.42 (12.73) | 2.67 (10.35)
  Day 10; n=10,6,6,6,6,6 | -0.10 (5.64) | -1.83 (10.52) | -4.33 (5.82) | -0.25 (7.62) | -3.33 (8.30) | -2.17 (7.82)
  Day 11; n=10,6,6,6,6,6 | 1.45 (7.98) | -2.58 (10.12) | -1.75 (6.33) | 0.00 (6.75) | 0.42 (12.46) | -3.58 (7.01)
  Day 12; n=10,6,6,6,6,6 | -0.50 (5.48) | -1.17 (12.30) | -2.33 (8.68) | 0.17 (4.69) | 1.75 (10.11) | 3.25 (11.02)
  Day 13; n=10,6,6,6,6,6 | 2.45 (5.83) | 2.00 (9.70) | -0.08 (8.63) | 2.92 (11.59) | -2.25 (11.49) | -2.08 (9.58)
  Day 14, Pre-dose; n=10,6,6,6,6,6 | -2.35 (3.93) | 0.25 (10.12) | -1.50 (10.11) | -2.17 (7.81) | -0.17 (7.75) | 0.42 (4.89)
  Day 14, 4 Hours Post-dose; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Day 14, 4 Hours Post-dose; n=10,5,6,6,6,6 | 0.40 (5.00) | 0.90 (11.06) | -5.75 (4.26) | -2.58 (7.39) | 3.83 (9.11) | -0.08 (6.67)
  Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Day 15; n=10,5,6,6,6,6 | 0.85 (4.34) | 4.00 (5.28) | 6.17 (9.68) | 4.00 (6.57) | 5.58 (8.03) | 7.67 (6.05)
  Follow-up (Day 25); n=10,6,6,6,6,6 | 6.25 (8.77) | 0.00 (6.67) | 4.25 (4.41) | 10.58 (8.44) | 5.83 (13.14) | 6.92 (6.85)

18. Primary Outcome: Part A: Change From Baseline in Body Temperature in Cohort 1 and Cohort 3
Description: Body temperature of participants was measured at indicated time points in a supine position after 5 minutes rest. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Pre-dose on Day 1), Day 1 (1, 4, 12 Hours Post-dose), Day 2 and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Celsius
  Day 1; 1 Hour Post dose | -0.09 (0.29) | 0.00 (0.00) | -0.22 (0.43) | -0.15 (0.31) | -0.12 (0.34) | 0.00 (0.00) | -0.20 (0.24)
  Day 1; 4 Hours Post dose | -0.09 (0.29) | 0.00 (0.00) | -0.22 (0.43) | -0.15 (0.31) | -0.12 (0.34) | 0.00 (0.00) | -0.20 (0.24)
  Day 1; 12 Hours Post dose | -0.09 (0.29) | 0.00 (0.00) | -0.22 (0.43) | -0.15 (0.31) | -0.12 (0.34) | 0.00 (0.00) | -0.20 (0.24)
  Day 2 | -0.04 (0.38) | -0.13 (0.37) | -0.27 (0.28) | -0.30 (0.42) | -0.58 (0.30) | -0.22 (0.29) | 0.00 (0.25)
  Day 3 | -0.07 (0.41) | -0.18 (0.26) | -0.45 (0.58) | 0.00 (0.49) | -0.16 (0.59) | 0.10 (0.48) | 0.26 (0.48)

19. Primary Outcome: Part A: Change From Baseline in Body Temperature in Cohort 2
Description: as for outcome 18
Time Frame: Baseline (Pre-dose on Day 1), Day 1 (1, 4, 12 Hours Post-dose), Day 2 and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Celsius
  Day 1; 1 Hour Post dose | 0.00 (0.00) | -0.10 (0.00) | 0.00 (0.00) | 0.00 (0.47)
  Day 1; 4 Hours Post dose | 0.00 (0.00) | -0.10 (0.00) | 0.00 (0.00) | 0.00 (0.47)
  Day 1; 12 Hours Post dose | 0.00 (0.00) | -0.10 (0.00) | 0.00 (0.00) | 0.00 (0.47)
  Day 2 | -0.15 (0.07) | -0.15 (0.21) | -0.33 (0.73) | 0.03 (0.39)
  Day 3 | -0.20 (0.14) | -0.35 (0.07) | -0.10 (0.49) | -0.22 (0.56)

20. Primary Outcome: Part B: Change From Baseline in Body Temperature
Description: Body temperature of participants was measured at indicated time points in a supine position after 5 minutes rest. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Celsius
  Day 1; 4 Hours Post dose; n=10,6,6,6,6,6 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 2; n=10,6,6,6,6,6 | 0.05 (0.32) | -0.03 (0.37) | 0.05 (0.30) | -0.02 (0.43) | 0.13 (0.47) | -0.20 (0.39)
  Day 3; n=10,6,6,6,6,6 | 0.09 (0.55) | -0.10 (0.15) | 0.05 (0.49) | 0.45 (0.33) | 0.13 (0.52) | 0.03 (0.42)
  Day 4; n=10,6,6,6,6,6 | 0.07 (0.31) | -0.10 (0.36) | -0.07 (0.49) | 0.05 (0.20) | 0.07 (0.35) | 0.03 (0.36)
  Day 5; n=10,6,6,6,6,6 | 0.16 (0.32) | 0.18 (0.13) | 0.23 (0.38) | 0.05 (0.21) | 0.27 (0.38) | -0.45 (0.38)
  Day 6; n=10,6,6,6,6,6 | 0.17 (0.51) | 0.33 (0.28) | -0.05 (0.48) | 0.53 (0.21) | 0.13 (0.57) | 0.05 (0.49)
  Day 7, Pre-dose; n=10,6,6,6,6,6 | 0.18 (0.45) | 0.12 (0.30) | 0.08 (0.38) | 0.23 (0.18) | 0.02 (0.29) | -0.08 (0.42)
  Day 7, 4 Hours Post-dose; n=10,6,6,6,6,6 | 0.18 (0.45) | 0.12 (0.30) | 0.08 (0.38) | 0.23 (0.18) | 0.02 (0.29) | -0.08 (0.42)
  Day 8; n=10,6,6,6,6,6 | 0.17 (0.34) | -0.02 (0.34) | 0.40 (0.37) | 0.08 (0.56) | 0.02 (0.54) | -0.15 (0.61)
  Day 9; n=10,6,6,6,6,6 | 0.08 (0.40) | 0.15 (0.32) | 0.30 (0.23) | 0.15 (0.39) | 0.23 (0.45) | -0.20 (0.62)
  Day 10; n=10,6,6,6,6,6 | -0.07 (0.51) | 0.17 (0.26) | 0.08 (0.45) | -0.10 (0.49) | -0.48 (0.60) | -0.02 (0.32)
  Day 11; n=10,6,6,6,6,6 | -0.05 (0.47) | 0.05 (0.39) | -0.02 (0.38) | 0.07 (0.42) | 0.00 (0.50) | -0.02 (0.39)
  Day 12; n=10,6,6,6,6,6 | -0.04 (0.67) | 0.00 (0.39) | -0.23 (0.45) | 0.55 (0.26) | -0.07 (0.45) | -0.08 (0.41)
  Day 13; n=10,6,6,6,6,6 | -0.07 (0.42) | 0.03 (0.37) | 0.15 (0.48) | -0.08 (0.18) | 0.05 (0.38) | -0.12 (0.40)
  Day 14, Pre-dose; n=10,6,6,6,6,6 | 0.17 (0.45) | 0.48 (0.31) | 0.27 (0.44) | 0.25 (0.31) | -0.10 (0.31) | -0.12 (0.48)
  Day 14, 4 Hours Post-dose; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Day 14, 4 Hours Post-dose; n=10,5,6,6,6,6 | 0.17 (0.45) | 0.42 (0.29) | 0.27 (0.44) | 0.25 (0.31) | -0.10 (0.31) | -0.12 (0.48)
  Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Day 15; n=10,5,6,6,6,6 | 0.27 (0.35) | 0.10 (0.24) | 0.47 (0.46) | 0.30 (0.55) | 0.28 (0.47) | 0.03 (0.31)
  Follow-up (Day 25); n=10,6,5,6,6,6: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6
  Follow-up (Day 25); n=10,6,5,6,6,6 | 0.18 (0.58) | 0.17 (0.52) | 0.24 (0.61) | 0.68 (0.34) | 0.47 (0.32) | 0.08 (0.36)

21. Primary Outcome: Part A: Number of Participants With Different Stool Types Assessed Using Bristol Stool Form Scale (BSFS) in Cohort 1
Description: The BSFS describes 7 types of stool as following; Type 1-Separate hard lumps (hard to pass), Type 2-Sausage-shaped but lumpy, Type 3-Like a sausage but cracks on surface, Type 4-Like a sausage or snake, smooth and soft, Type 5- Soft blobs with clear cut edges, Type-6 Fluffy pieces with ragged edges, a mushy stool, and Type 7-Watery, no solid pieces (entirely liquid). BSFS was used by the participants during the study to capture the quality of stool using a 7-point scale ranging from Type 1=separate hard lumps like nuts (difficult to pass) to 7= watery, no solid pieces (entirely liquid).
Time Frame: Up to 64 days in Cohort 1
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 5
Participants
  Type 1 | 0 | 0 | 0 | 1 | 0
  Type 2 | 3 | 3 | 2 | 0 | 0
  Type 3 | 3 | 1 | 2 | 3 | 1
  Type 4 | 1 | 1 | 2 | 1 | 3
  Type 5 | 4 | 3 | 2 | 3 | 1
  Type 6 | 3 | 0 | 2 | 2 | 1
  Type 7 | 0 | 0 | 1 | 0 | 0

22. Primary Outcome: Part A: Number of Participants With Different Stool Types Assessed Using BSFS in Cohort 2
Description: as for outcome 21
Time Frame: Up to 30 days in Cohort 2
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Participants
  Type 1 | 0 | 0 | 0 | 0
  Type 2 | 0 | 0 | 3 | 1
  Type 3 | 1 | 1 | 2 | 3
  Type 4 | 1 | 1 | 3 | 1
  Type 5 | 0 | 0 | 1 | 0
  Type 6 | 0 | 0 | 0 | 1
  Type 7 | 0 | 0 | 0 | 0

23. Primary Outcome: Part A: Number of Participants With Different Stool Types Assessed Using BSFS in Cohort 3
Description: as for outcome 21
Time Frame: Up to 30 days in Cohort 3
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 3: Placebo | Part A: Cohort 3: GSK3352589 150 mg | Part A: Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 4 | 6 | 5
Participants
  Type 1 | 0 | 0 | 1
  Type 2 | 0 | 1 | 0
  Type 3 | 2 | 4 | 3
  Type 4 | 2 | 5 | 5
  Type 5 | 0 | 3 | 2
  Type 6 | 1 | 0 | 0
  Type 7 | 0 | 0 | 0

24. Primary Outcome: Part B: Average BSFS at Indicated Time Points
Description: as for outcome 21
Time Frame: Day -1, Days 1-3, Days 4-7, Days 1-7, Days 8-14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Units on a scale
  Day -1; n=7,4, 6,6,4,5: number analyzed (Participants) | 7 | 4 | 6 | 6 | 4 | 5
  Day -1; n=7,4, 6,6,4,5 | 3.17 (1.30) | 3.88 (0.63) | 3.92 (0.49) | 3.92 (1.43) | 4.13 (1.03) | 4.30 (0.84)
  Days 1-3; n=10,6,6,6,6,6 | 3.93 (1.14) | 3.55 (1.57) | 3.97 (1.06) | 3.62 (0.71) | 3.75 (1.33) | 3.37 (0.91)
  Days 4-7;n=9,6,6,6,6,6: number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 6
  Days 4-7;n=9,6,6,6,6,6 | 4.32 (1.14) | 3.78 (1.30) | 3.68 (1.14) | 3.37 (0.47) | 3.85 (0.95) | 3.45 (0.34)
  Days 1-7;n=10,6,6,6,6,6 | 4.14 (0.99) | 3.75 (1.36) | 3.77 (0.86) | 3.48 (0.50) | 3.78 (1.08) | 3.38 (0.34)
  Days 8-14;n=10,6,6,6,6,6 | 4.12 (0.97) | 3.63 (1.12) | 3.93 (0.77) | 3.10 (0.63) | 3.63 (1.29) | 3.48 (0.48)

25. Primary Outcome: Part A: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, Leukocytes in Cohort 1 and Cohort 3
Description: Blood samples were collected for analysis of hematology parameters including Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, and Leukocytes. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1) and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
10^9 cells per liter
  Basophils; Day 3 | 0.01 (0.05) | 0.00 (0.06) | 0.02 (0.04) | 0.00 (0.06) | 0.04 (0.05) | -0.03 (0.05) | -0.05 (0.05)
  Eosinophils; Day 3 | 0.02 (0.06) | 0.02 (0.08) | 0.05 (0.14) | -0.03 (0.05) | 0.02 (0.05) | 0.02 (0.04) | 0.04 (0.05)
  Lymphocytes; Day 3 | -0.37 (0.40) | -0.10 (0.40) | -0.32 (0.46) | -0.43 (0.36) | -0.50 (0.34) | 0.03 (0.31) | -0.16 (0.29)
  Monocytes; Day 3 | -0.05 (0.12) | -0.08 (0.10) | -0.13 (0.08) | -0.08 (0.12) | -0.04 (0.21) | 0.03 (0.08) | 0.02 (0.04)
  Neutrophils; Day 3 | -0.66 (1.05) | -0.73 (1.06) | -0.60 (1.55) | -0.23 (0.70) | -0.16 (2.76) | -0.60 (0.85) | -0.36 (0.90)
  Platelets; Day 3 | -15.0 (34.6) | -4.8 (34.1) | -22.5 (45.6) | 2.2 (32.4) | -8.0 (43.7) | -23.3 (13.9) | -46.6 (36.5)
  Leukocytes ;Day 3 | -1.01 (1.06) | -0.88 (0.95) | -0.95 (1.33) | -0.82 (0.80) | -0.58 (2.64) | -0.53 (0.94) | -0.52 (0.94)

26. Primary Outcome: Part A: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, Leukocytes in Cohort 2
Description: as for outcome 25
Time Frame: Baseline (Day -1) and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
10^9 cells per liter
  Basophils; Day 3 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.02 (0.04)
  Eosinophils; Day 3 | 0.05 (0.08) | 0.05 (0.07) | 0.00 (0.06) | 0.03 (0.06)
  Lymphocytes; Day 3 | 0.10 (0.14) | 0.10 (0.14) | 0.25 (0.65) | 0.12 (0.58)
  Monocytes; Day 3 | -0.05 (0.07) | -0.05 (0.07) | -0.02 (0.15) | -0.08 (0.10)
  Neutrophils; Day 3 | -1.00 (0.42) | -0.85 (0.35) | -1.25 (1.97) | -1.73 (1.84)
  Platelets; Day 3 | -7.0 (11.3) | -45.0 (26.9) | -7.2 (5.9) | -29.2 (27.0)
  Leukocytes ;Day 3 | -0.90 (0.57) | -0.75 (0.35) | -1.00 (2.44) | -1.68 (2.30)

27. Primary Outcome: Part B: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, Leukocytes
Description: Blood samples were collected for analysis of hematology parameters including Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, and Leukocytes. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), Day 7, Day 15 and Follow-up (Day 25)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
10^9 cells per liter
  Basophils; Day 7;n=10, 6,6,6,6,6 | 0.03 (0.06) | 0.00 (0.06) | 0.05 (0.05) | 0.03 (0.05) | 0.02 (0.04) | 0.02 (0.04)
  Basophils; Day 15;n=10, 5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Basophils; Day 15;n=10, 5,6,6,6,6 | 0.03 (0.06) | 0.04 (0.05) | 0.05 (0.05) | 0.05 (0.05) | 0.03 (0.05) | 0.02 (0.04)
  Basophils; Follow-up (Day 25) ; n=10, 6,6,6,6,6 | 0.05 (0.05) | 0.00 (0.06) | 0.06 (0.05) | 0.05 (0.05) | 0.02 (0.07) | 0.00 (0.00)
  Eosinophils; Day 7;n=10, 6,6,6,6,6 | 0.01 (0.09) | 0.03 (0.05) | -0.02 (0.04) | 0.03 (0.08) | 0.05 (0.05) | 0.04 (0.08)
  Eosinophils, Day 15;n=10, 5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Eosinophils, Day 15;n=10, 5,6,6,6,6 | 0.02 (0.10) | 0.04 (0.11) | 0.02 (0.04) | 0.03 (0.08) | 0.05 (0.05) | -0.03 (0.08)
  Eosinophils; Follow-up (Day 25); n=10, 6,6,6,6,6 | 0.01 (0.09) | 0.05 (0.09) | 0.04 (0.05) | 0.03 (0.10) | 0.05 (0.08) | -0.03 (0.11)
  Lymphocytes; Day 7 ;n=10, 6,6,6,6,6 | -0.09 (0.35) | -0.35 (0.26) | -0.18 (0.24) | -0.10 (0.30) | 0.23 (0.19) | -0.22 (0.40)
  Lymphocytes; Day 15; n=10, 5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Lymphocytes; Day 15; n=10, 5,6,6,6,6 | 0.04 (0.32) | 0.02 (0.22) | 0.10 (0.20) | -0.05 (0.36) | 0.40 (0.25) | -0.10 (0.19)
  Lymphocytes; Follow-up (Day 25); n=10, 6,6,6,6,6 | 0.14 (0.25) | -0.12 (0.33) | 0.25 (0.35) | 0.00 (0.13) | 0.07 (0.23) | -0.32 (0.17)
  Monocytes; Day 7;n=10, 6,6,6,6,6 | -0.03 (0.09) | -0.03 (0.05) | -0.08 (0.12) | -0.10 (0.06) | 0.05 (0.10) | 0.02 (0.08)
  Monocytes; Day 15;n=10, 5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Monocytes; Day 15;n=10, 5,6,6,6,6 | -0.09 (0.11) | -0.02 (0.04) | -0.02 (0.08) | -0.10 (0.09) | 0.05 (0.05) | -0.07 (0.08)
  Monocytes; Follow-up (Day 25); n=10, 6,6,6,6,6 | -0.04 (0.12) | -0.05 (0.10) | 0.03 (0.08) | -0.10 (0.06) | 0.17 (0.27) | -0.07 (0.10)
  Neutrophils; Day 7;n=10, 6,6,6,6,6 | -0.08 (1.05) | 0.05 (0.57) | -0.42 (0.34) | -0.65 (0.98) | -0.82 (0.79) | -0.88 (0.57)
  Neutrophils; Day 15;n=10, 5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Neutrophils; Day 15;n=10, 5,6,6,6,6 | -0.31 (0.74) | -0.02 (0.39) | -0.22 (0.77) | -0.72 (0.87) | -0.58 (0.50) | -0.95 (0.75)
  Neutrophils; Follow-up (Day 25); n=10, 6,6,6,6,6 | -0.55 (0.94) | 0.05 (0.42) | 0.07 (0.66) | -0.37 (1.33) | 0.73 (3.34) | -0.58 (1.05)
  Platelets; Day 7;n=10, 6,6,6,6,6 | 10.4 (25.0) | 9.7 (21.9) | 8.3 (20.8) | 26.7 (12.1) | -11.0 (12.1) | 4.5 (21.1)
  Platelets; Day 15;n=10, 5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Platelets; Day 15;n=10, 5,6,6,6,6 | 12.3 (28.5) | 24.2 (26.7) | -3.0 (23.9) | 3.7 (16.6) | 7.3 (25.5) | 7.5 (21.3)
  Platelets; Follow-up (Day 25); n=10, 6,6,6,6,6 | 17.5 (34.5) | 37.3 (24.3) | 26.2 (24.2) | 27.3 (37.0) | 2.5 (20.9) | 2.5 (9.0)
  Leukocytes; Day 7;n=10, 6,6,6,6,6 | -0.18 (1.13) | -0.32 (0.52) | -0.65 (0.60) | -0.82 (1.00) | -0.53 (0.92) | -1.08 (0.67)
  Leukocytes ;Day 15;n=10, 5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Leukocytes ;Day 15;n=10, 5,6,6,6,6 | -0.32 (0.79) | 0.10 (0.47) | -0.13 (0.76) | -0.82 (0.85) | -0.08 (0.45) | -1.10 (0.62)
  Leukocytes; Follow-up (Day 25); n=10, 6,6,6,6,6 | -0.39 (0.72) | -0.12 (0.59) | 0.43 (0.88) | -0.45 (1.24) | 0.98 (3.38) | -1.00 (1.01)

28. Primary Outcome: Part A: Change From Baseline in Erythrocytes in Cohort 1 and 3
Description: Blood samples were collected for analysis of hematology parameters including Erythrocytes. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1) and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
10^12 cells per liter | 0.029 (0.260) | 0.275 (0.321) | -0.073 (0.310) | 0.112 (0.390) | 0.120 (0.373) | 0.063 (0.094) | -0.132 (0.132)

29. Primary Outcome: Part A: Change From Baseline in Erythrocytes in Cohort 2
Description: as for outcome 28
Time Frame: Baseline (Day -1) and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
10^12 cells per liter | 0.110 (0.156) | 0.150 (0.269) | 0.167 (0.118) | 0.042 (0.157)

30. Primary Outcome: Part B: Change From Baseline in Erythrocytes
Description: Blood samples were collected for analysis of hematology parameters including Erythrocytes. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), Day 7, Day 15 and Follow-up (Day 25)
Population: Safety population. Only those participants with data available at specified time point were analyzed (reported by n=X in category titles).
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
10^12 cells per liter
  Day 7; n=10,6,6,6,6,6 | 0.081 (0.250) | 0.208 (0.119) | 0.033 (0.060) | 0.230 (0.145) | -0.183 (0.183) | -0.023 (0.251)
  Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Day 15; n=10,5,6,6,6,6 | 0.175 (0.258) | 0.334 (0.235) | 0.270 (0.190) | 0.302 (0.179) | 0.162 (0.252) | 0.082 (0.275)
  Follow-up (Day 25); n=10,6,6,6,6,6 | 0.075 (0.355) | 0.287 (0.256) | 0.155 (0.182) | 0.158 (0.239) | -0.195 (0.165) | -0.227 (0.157)

31. Primary Outcome: Part A: Change From Baseline in Hemoglobin in Cohort 1 and 3
Description: Blood samples were collected for analysis of hematology parameters including hemoglobin. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1) and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Grams per liter | 0.0 (8.3) | 6.2 (9.0) | -2.5 (9.3) | 2.0 (9.0) | -0.8 (8.8) | 2.2 (4.3) | -1.2 (4.3)

32. Primary Outcome: Part A: Change From Baseline in Hemoglobin in Cohort 2
Description: as for outcome 31
Time Frame: Baseline (Day -1) and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Grams per liter | 4.0 (2.8) | 5.5 (9.2) | 5.8 (3.3) | 2.3 (3.8)

33. Primary Outcome: Part B: Change From Baseline in Hemoglobin
Description: Blood samples were collected for analysis of hematology parameters including hemoglobin. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), Day 7, Day 15 and Follow-up (Day 25)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Grams per liter
  Day 7; n=10,6,6,6,6,6 | -1.8 (6.5) | 1.8 (4.5) | -5.3 (2.0) | 0.7 (4.1) | -6.7 (4.3) | 0.0 (6.9)
  Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Day 15; n=10,5,6,6,6,6 | 1.4 (8.7) | 6.4 (6.7) | 1.3 (5.6) | 3.7 (5.4) | 2.2 (4.9) | 3.7 (6.4)
  Follow-up (Day 25); n=10,6,6,6,6,6 | -1.3 (10.4) | 4.3 (7.1) | -1.8 (5.6) | -0.3 (5.9) | -3.5 (4.5) | -3.0 (4.6)

34. Primary Outcome: Part A: Change From Baseline in Erythrocyte Mean Corpuscular Volume (MCV) in Cohort 1 and Cohort 3
Description: Blood samples were collected for analysis of hematology parameters including Erythrocyte MCV. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1) and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Femtoliter | 0.9 (1.1) | 0.2 (1.5) | 1.5 (0.8) | 1.7 (1.2) | 1.6 (1.1) | 0.8 (0.8) | 1.0 (1.6)

35. Primary Outcome: Part A: Change From Baseline in Erythrocyte MCV in Cohort 2
Description: as for outcome 34
Time Frame: Baseline (Day -1) and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Femtoliter | -2.0 (1.4) | -2.0 (1.4) | 1.5 (3.0) | 0.7 (2.6)

36. Primary Outcome: Part B: Change From Baseline in Erythrocyte MCV
Description: Blood samples were collected for analysis of hematology parameters including Erythrocyte MCV. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), Day 7, Day 15 and Follow-up (Day 25)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Femtoliter
  Day 7; n=10,6,6,6,6,6 | -1.4 (1.6) | 0.2 (1.2) | -2.7 (1.8) | -0.2 (0.8) | 0.2 (1.2) | -1.3 (1.5)
  Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Day 15; n=10,5,6,6,6,6 | -1.0 (1.2) | 0.2 (1.9) | -2.2 (1.7) | -0.3 (1.4) | 0.8 (1.2) | -0.8 (1.9)
  Follow-up (Day 25); n=10,6,6,6,6,6 | -0.5 (1.9) | 0.0 (1.4) | -1.5 (1.9) | 0.3 (0.8) | 1.8 (0.4) | 0.0 (0.9)

37. Primary Outcome: Part A: Change From Baseline in Erythorocyte Mean Corpuscular Hemoglobin (MCH) in Cohort 1 and 3
Description: Blood samples were collected for analysis of hematology parameters including Erythorocyte MCH. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1) and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Picogram | -0.19 (0.71) | -0.37 (0.47) | -0.13 (0.40) | -0.25 (0.66) | -0.84 (0.52) | 0.08 (0.35) | 0.54 (0.43)

38. Primary Outcome: Part A: Change From Baseline in Erythrocyte MCH in Cohort 2
Description: as for outcome 37
Time Frame: Baseline (Day -1) and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Picogram | 0.20 (0.28) | 0.20 (0.28) | 0.20 (0.37) | 0.27 (0.23)

39. Primary Outcome: Part B: Change From Baseline in Erythrocyte MCH
Description: Blood samples were collected for analysis of hematology parameters including Erythorocyte MCH. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), Day 7, Day 15 and Follow-up (Day 25)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Picogram
  Day 7; n=10,6,6,6,6,6 | -0.87 (0.55) | -0.87 (0.37) | -1.25 (0.40) | -1.13 (0.21) | -0.28 (0.34) | 0.13 (0.85)
  Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Day 15; n=10,5,6,6,6,6 | -0.77 (0.72) | -0.70 (0.37) | -1.33 (0.14) | -0.95 (0.38) | -0.50 (0.46) | 0.23 (0.81)
  Follow-up (Day 25); n=10,6,6,6,6,6 | -0.72 (0.57) | -0.78 (0.58) | -1.30 (0.25) | -0.98 (0.26) | 0.47 (0.39) | 0.77 (0.54)

40. Primary Outcome: Part A: Change From Baseline in Hematocrit in Cohort 1 and 3
Description: Blood samples were collected for analysis of hematology parameters including Hematocrit. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1) and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Proportion of red blood cells in blood | 0.007 (0.021) | 0.025 (0.027) | 0.002 (0.029) | 0.017 (0.031) | 0.018 (0.026) | 0.007 (0.008) | -0.008 (0.015)

41. Primary Outcome: Part A: Change From Baseline in Hematocrit in Cohort 2
Description: as for outcome 40
Time Frame: Baseline (Day -1) and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Proportion of red blood cells in blood | 0.005 (0.021) | 0.010 (0.028) | 0.023 (0.020) | 0.008 (0.015)

42. Primary Outcome: Part B: Change From Baseline in Hematocrit
Description: Blood samples were collected for analysis of hematology parameters including Hematocrit. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), Day 7, Day 15 and Follow-up (Day 25)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Proportion of red blood cells in blood
  Day 7; n=10,6,6,6,6,6 | 0.000 (0.029) | 0.018 (0.010) | -0.012 (0.012) | 0.018 (0.013) | -0.017 (0.014) | -0.007 (0.020)
  Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Day 15; n=10,5,6,6,6,6 | 0.009 (0.025) | 0.030 (0.025) | 0.015 (0.018) | 0.025 (0.016) | 0.017 (0.019) | 0.005 (0.026)
  Follow-up (Day 25); n=10,6,6,6,6,6 | 0.005 (0.032) | 0.025 (0.021) | 0.005 (0.016) | 0.017 (0.020) | -0.008 (0.015) | -0.020 (0.017)

43. Primary Outcome: Part A: Change From Baseline in Alanine Aminotransferase (ALT),Aspartate Aminotransferase (AST), Alkaline Phosphatase (Alk Phos) in Cohort 1 and 3
Description: Blood samples were collected for analysis of clinical chemistry parameters including ALT, AST and Alk Phos. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1) and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Units per liter
  ALT; Day 3 | 5.0 (27.1) | -1.8 (15.0) | -6.2 (12.4) | -1.2 (14.2) | -7.2 (15.6) | 6.0 (3.2) | 8.0 (9.3)
  AST; Day 3 | 1.3 (10.3) | 1.0 (8.1) | -0.2 (5.3) | -0.2 (5.3) | -1.8 (4.7) | -5.0 (5.2) | -3.4 (5.5)
  Alk Phos; Day 3 | -5.9 (11.7) | -7.3 (7.5) | -9.2 (8.9) | -10.5 (8.7) | -17.0 (6.6) | 0.2 (6.5) | -3.6 (8.2)

44. Primary Outcome: Part A: Change From Baseline in ALT, AST and Alk Phos in Cohort 2
Description: as for outcome 43
Time Frame: Baseline (Day -1) and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Units per liter
  ALT; Day 3 | -1.5 (0.7) | -0.5 (2.1) | 0.2 (1.5) | -2.3 (5.6)
  AST; Day 3 | -4.5 (0.7) | -1.5 (2.1) | -4.5 (3.3) | -4.3 (4.2)
  Alk Phos; Day 3 | -6.0 (5.7) | -10.0 (4.2) | 0.8 (5.8) | -2.0 (4.6)

45. Primary Outcome: Part B: Change From Baseline in ALT, AST and Alk Phos
Description: Blood samples were collected for analysis of hematology parameters including ALT, AST and Alk Phos. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), Day 7, Day 15 and Follow-up (Day 25)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Units per liter
  ALT; Day 7; n=10,6,6,6,6,6 | -4.8 (10.9) | -7.7 (5.9) | -6.2 (6.0) | 2.3 (5.5) | -0.8 (2.8) | -0.3 (2.4)
  ALT; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  ALT; Day 15; n=10,5,6,6,6,6 | -1.3 (11.9) | -8.2 (4.7) | -5.3 (8.1) | -3.8 (6.7) | -0.7 (4.1) | -0.8 (3.8)
  ALT; Follow-up (Day 25); n=10,6,6,6,6,6 | -5.3 (9.0) | -7.8 (5.3) | -9.3 (7.7) | -1.0 (6.8) | 0.3 (7.6) | -2.3 (3.3)
  AST ; Day 7; n=10,6,6,6,6,6 | 2.8 (18.5) | 0.3 (4.5) | 3.5 (7.7) | 7.7 (6.1) | 3.0 (10.4) | 0.7 (3.6)
  AST; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  AST; Day 15; n=10,5,6,6,6,6 | 0.5 (5.3) | -1.6 (4.2) | 3.2 (6.7) | 0.5 (3.3) | -0.8 (2.9) | -0.3 (3.9)
  AST; Follow-up (Day 25); n=10,6,6,6,6,6 | -0.4 (4.0) | -0.2 (5.5) | 1.7 (5.1) | 7.7 (16.0) | 1.2 (4.4) | -1.2 (4.6)
  Alk Phos; Day 7; n=10,6,6,6,6,6 | -6.7 (4.4) | -7.3 (9.4) | -8.7 (4.9) | -2.8 (6.6) | -10.5 (5.6) | -1.8 (6.1)
  Alk Phos ; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Alk Phos ; Day 15; n=10,5,6,6,6,6 | -4.3 (5.9) | -1.4 (3.6) | -5.3 (6.5) | -0.5 (7.5) | -4.8 (6.8) | 0.7 (6.7)
  Alk Phos ; Follow-up (Day 25); n=10,6,6,6,6,6 | -3.5 (8.0) | -7.8 (17.8) | -6.2 (8.8) | 1.2 (12.4) | -0.7 (7.1) | 0.7 (3.0)

46. Primary Outcome: Part A: Change From Baseline in Bilirubin, Creatinine, Direct Bilirubin in Cohort 1 and 3
Description: Blood samples were collected for analysis of clinical chemistry parameters including bilirubin, creatinine, direct bilirubin. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1) and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Micromoles per liter
  Bilirubin; Day 3 | 1.2 (3.3) | 1.0 (4.2) | 1.2 (3.0) | 2.2 (1.9) | 1.6 (3.4) | -0.7 (4.4) | 2.2 (3.7)
  Creatinine; Day 3 | -0.7 (7.0) | -2.5 (5.3) | -2.3 (8.5) | 1.7 (8.6) | 0.4 (11.1) | 1.5 (5.0) | -3.0 (13.4)
  Direct bilirubin; Day 3 | 0.80 (1.49) | 0.85 (1.86) | 0.52 (0.74) | 1.38 (0.90) | 1.58 (1.00) | -1.15 (1.84) | -0.14 (1.00)

47. Primary Outcome: Part A: Change From Baseline in Bilirubin, Creatinine, Direct Bilirubin in Cohort 2
Description: Blood samples were collected for analysis of clinical chemistry parameters including bilirubin, creatinine, and direct bilirubin. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Micromoles per liter
  Bilirubin; Day 3 | 3.5 (2.1) | 2.0 (1.4) | 1.5 (3.4) | -0.7 (4.3)
  Creatinine; Day 3 | -8.5 (7.8) | -8.0 (8.5) | -2.2 (4.6) | -5.3 (4.3)
  Direct bilirubin; Day 3 | 0.65 (0.35) | 0.50 (0.00) | 0.38 (0.87) | -0.10 (1.33)

48. Primary Outcome: Part B: Change From Baseline in Bilirubin, Creatinine, Direct Bilirubin
Description: Blood samples were collected for analysis of hematology parameters including bilirubin, creatinine, and direct bilirubin. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), Day 7, Day 15 and Follow-up (Day 25)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Micromoles per liter
  Bilirubin; Day 7; n=10,6,6,6,6,6 | 2.4 (1.7) | 2.5 (1.9) | 3.2 (2.8) | 2.0 (1.7) | 2.0 (2.8) | 2.5 (4.2)
  Bilirubin; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Bilirubin; Day 15; n=10,5,6,6,6,6 | 1.9 (2.0) | 1.0 (2.4) | 2.5 (1.5) | 1.5 (1.6) | 2.3 (2.9) | 2.0 (3.4)
  Bilirubin; Follow-up (Day 25);n=10,6,6,6,6,6 | 1.2 (1.6) | 0.5 (4.4) | 2.5 (2.2) | 1.8 (3.5) | 0.3 (4.4) | 0.8 (3.8)
  Creatinine ; Day 7; n=10,6,6,6,6,6 | 0.2 (6.5) | -5.5 (14.0) | -1.3 (15.7) | -3.3 (7.3) | -13.0 (9.2) | -1.0 (6.7)
  Creatinine; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Creatinine; Day 15; n=10,5,6,6,6,6 | -3.0 (5.3) | 2.2 (12.7) | -1.0 (15.3) | -1.0 (7.8) | -9.2 (13.2) | -2.7 (4.5)
  Creatinine; Follow-up (Day 25); n=10,6,6,6,6,6 | 3.4 (6.9) | -1.0 (16.6) | 0.8 (15.0) | 0.5 (7.1) | -4.0 (11.3) | -1.3 (5.2)
  Direct bilirubin ; Day 7; n=10,6,6,6,6,6 | 1.31 (0.43) | 1.30 (0.59) | 1.32 (1.22) | 1.22 (0.64) | 0.48 (1.15) | 0.63 (1.53)
  Direct bilirubin ; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Direct bilirubin ; Day 15; n=10,5,6,6,6,6 | 1.00 (0.67) | 1.10 (0.54) | 0.73 (0.81) | 1.73 (0.46) | 0.73 (1.17) | 0.25 (1.51)
  Direct bilirubin; Follow-up(Day 25);n=10,6,6,6,6,6 | 1.06 (0.62) | 1.10 (1.05) | 0.95 (0.87) | 1.78 (1.06) | -0.12 (1.42) | 0.48 (1.23)

49. Primary Outcome: Part A: Change From Baseline in Calcium, Glucose, Potassium, Sodium, Urea in Cohort 1 and 3
Description: Blood samples were collected for analysis of clinical chemistry parameters including Calcium, Glucose, Potassium, Sodium, Urea. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1) and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Millimoles per liter
  Calcium; Day 3 | -0.049 (0.108) | -0.005 (0.134) | -0.075 (0.107) | -0.060 (0.145) | -0.054 (0.152) | -0.063 (0.038) | -0.124 (0.067)
  Glucose; Day 3 | 0.01 (0.69) | -0.03 (0.27) | 0.25 (0.82) | 0.22 (0.36) | -0.32 (1.32) | -0.23 (0.64) | 0.22 (0.94)
  Potassium; Day 3 | -0.04 (0.28) | 0.05 (0.30) | 0.13 (0.35) | 0.10 (0.23) | -0.08 (0.16) | -0.03 (0.27) | 0.16 (0.17)
  Sodium; Day 3 | -2.5 (2.2) | -2.7 (2.1) | -2.3 (3.0) | -1.8 (1.5) | -2.0 (1.9) | -1.0 (2.6) | 1.0 (1.0)
  Urea; Day 3 | -0.43 (1.11) | -0.62 (0.74) | -0.68 (1.39) | -0.13 (1.22) | -0.14 (0.80) | -0.55 (1.20) | -0.48 (0.57)

50. Primary Outcome: Part A: Change From Baseline in Calcium, Glucose, Potassium, Sodium, Urea in Cohort 2
Description: as for outcome 49
Time Frame: Baseline (Day -1) and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Millimoles per liter
  Calcium; Day 3 | -0.075 (0.078) | -0.110 (0.071) | 0.022 (0.120) | -0.037 (0.105)
  Glucose; Day 3 | 0.35 (0.21) | 0.30 (0.14) | -0.45 (0.49) | -0.55 (0.52)
  Potassium; Day 3 | 0.05 (0.07) | 0.05 (0.07) | -0.17 (0.27) | -0.13 (0.29)
  Sodium; Day 3 | 0.0 (0.0) | 1.0 (1.4) | 0.7 (1.2) | 0.5 (2.2)
  Urea; Day 3 | -1.30 (0.14) | -1.00 (0.57) | 0.37 (1.15) | -0.03 (1.32)

51. Primary Outcome: Part B: Change From Baseline in Calcium, Glucose, Potassium, Sodium, Urea
Description: Blood samples were collected for analysis of hematology parameters including Calcium, Glucose, Potassium, Sodium, Urea. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), Day 7, Day 15 and Follow-up (Day 25)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Millimoles per liter
  Calcium; Day 7; n=10,6,6,6,6,6 | -0.001 (0.086) | 0.040 (0.065) | 0.108 (0.027) | 0.050 (0.055) | -0.045 (0.106) | -0.035 (0.100)
  Calcium; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Calcium; Day 15; n=10,5,6,6,6,6 | 0.026 (0.142) | 0.124 (0.093) | 0.167 (0.044) | 0.073 (0.026) | 0.052 (0.098) | -0.032 (0.138)
  Calcium; Follow-up (Day 25); n=10,6,6,6,6,6 | 0.049 (0.177) | 0.160 (0.067) | 0.157 (0.061) | 0.100 (0.059) | -0.023 (0.080) | -0.005 (0.099)
  Glucose; Day 7; n=10,6,6,6,6,6 | -0.16 (0.80) | -0.78 (0.69) | -0.05 (0.45) | -0.17 (0.46) | -0.47 (0.46) | -0.33 (0.47)
  Glucose; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Glucose; Day 15; n=10,5,6,6,6,6 | -0.37 (0.81) | -0.70 (0.62) | -0.17 (0.52) | -0.72 (0.35) | -1.02 (0.55) | -0.40 (0.40)
  Glucose; Follow-up (Day 25); n=10,6,6,6,6,6 | 0.21 (0.96) | -0.03 (1.00) | -0.30 (0.67) | -0.08 (0.38) | -0.08 (1.21) | -0.12 (0.98)
  Potassium; Day 7; n=10,6,6,6,6,6 | 0.22 (0.64) | -0.17 (0.39) | 0.38 (0.42) | 0.57 (0.21) | 0.15 (0.74) | -0.05 (0.23)
  Potassium; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Potassium; Day 15; n=10,5,6,6,6,6 | -0.06 (0.33) | -0.06 (0.54) | 0.47 (0.37) | 0.18 (0.15) | -0.02 (0.31) | 0.07 (0.36)
  Potassium; Follow-up (Day 25); n=10,6,6,6,6,6 | 0.04 (0.41) | 0.03 (0.43) | 0.23 (0.23) | -0.07 (0.41) | -0.10 (0.32) | 0.00 (0.28)
  Sodium; Day 7; n=10,6,6,6,6,6 | -1.8 (2.7) | -2.7 (2.0) | -0.3 (1.6) | -0.8 (2.6) | -2.3 (3.0) | -0.3 (2.1)
  Sodium; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Sodium; Day 15; n=10,5,6,6,6,6 | -1.8 (2.7) | -2.0 (2.9) | -0.5 (0.8) | 1.0 (2.7) | 1.8 (3.4) | 0.3 (2.3)
  Sodium; Follow-up (Day 25); n=10,6,6,6,6,6 | -1.6 (2.8) | -2.3 (2.4) | -0.5 (1.2) | 0.8 (2.2) | 0.7 (3.3) | 0.2 (0.8)
  Urea; Day 7; n=10,6,6,6,6,6 | -0.84 (0.88) | -0.52 (0.75) | -2.58 (2.10) | -0.43 (0.42) | -1.18 (1.28) | -0.20 (0.75)
  Urea; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Urea; Day 15; n=10,5,6,6,6,6 | -1.56 (1.04) | -0.88 (0.79) | -2.82 (2.01) | -1.17 (0.31) | -1.40 (1.21) | -1.25 (0.78)
  Urea; Follow-up (Day 25); n=10,6,6,6,6,6 | 0.48 (1.04) | 0.50 (1.69) | -0.27 (0.91) | -0.40 (1.39) | -1.10 (1.67) | -0.03 (1.03)

52. Primary Outcome: Part A: Change From Baseline in Albumin and Total Protein in Cohort 1 and 3
Description: Blood samples were collected for analysis of clinical chemistry parameters including albumin, and total protein. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1) and Day 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Grams per liter
  Albumin; Day 3 | -3.1 (3.5) | -1.8 (4.8) | -3.5 (4.3) | -3.2 (3.1) | -4.8 (3.8) | -2.8 (2.2) | -3.8 (2.8)
  Total Protein; Day 3 | -3.5 (5.8) | -2.5 (6.9) | -5.0 (7.4) | -3.3 (5.3) | -6.2 (7.1) | -2.0 (3.6) | -2.6 (3.4)

53. Primary Outcome: Part A: Change From Baseline in Albumin and Total Protein in Cohort 2
Description: Blood samples were collected for analysis of clinical chemistry parameters including albumin and total protein. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period 1 (or the first available Dosing Period if Dosing Period 1 is unavailable). Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Grams per liter
  Albumin; Day 3 | -1.0 (0.0) | -2.0 (0.0) | -1.2 (2.7) | -1.7 (2.9)
  Total Protein; Day 3 | -2.5 (0.7) | -4.5 (2.1) | -1.5 (5.1) | -3.8 (2.9)

54. Primary Outcome: Part B: Change From Baseline in Albumin, Total Protein
Description: Blood samples were collected for analysis of hematology parameters including albumin and total protein. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), Day 7, Day 15 and Follow-up (Day 25)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Grams per liter
  Albumin; Day 7; n=10,6,6,6,6,6 | -2.5 (1.9) | -2.3 (1.4) | -2.2 (0.8) | -3.3 (1.9) | -3.7 (1.4) | -0.8 (3.1)
  Albumin; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Albumin; Day 15; n=10,5,6,6,6,6 | -2.2 (2.6) | -0.4 (2.2) | 0.2 (1.5) | -2.5 (2.3) | -0.7 (1.2) | -1.0 (3.5)
  Albumin; Follow-up (Day 25);n=10,6,6,6,6,6 | -0.7 (2.5) | -0.3 (3.3) | 1.2 (1.0) | 0.2 (3.6) | -1.7 (1.4) | -0.5 (2.9)
  Total Protein; Day 7; n=10,6,6,6,6,6 | -3.0 (3.2) | -2.5 (2.1) | -4.0 (2.3) | -1.8 (2.1) | -4.5 (2.3) | -1.2 (4.5)
  Total Protein; Day 15; n=10,5,6,6,6,6: number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
  Total Protein; Day 15; n=10,5,6,6,6,6 | -2.9 (3.7) | 0.2 (4.1) | -0.3 (3.1) | -1.3 (3.0) | -1.0 (2.8) | 0.2 (5.4)
  Total Protein;Follow-up (Day 25); n=10,6,6,6,6,6 | -1.4 (4.8) | 0.8 (4.9) | 0.5 (1.9) | 2.0 (4.4) | -2.2 (2.5) | -1.3 (4.0)

55. Primary Outcome: Part A: Number of Participants With Abnormal Findings for Urine Parameters in Cohort 1 and Cohort 3
Description: Urine samples were collected from participants for analysis of specific gravity of urine. Urine parameters including bilirubin, glucose, ketones, leukocyte esterase, nitrite, occult blood, potential of hydrogen (pH), protein, specific gravity and Urobilinogen were analyzed by dipstick method. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug in Dosing Period
  1 (or the first available Dosing Period if Dosing Period 1 is unavailable).
Time Frame: Baseline (Day-1) and Day 3
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 and 3: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A:Cohort 3: GSK3352589 150 mg | Part A:Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 5 | 6 | 5
Participants
  Bilirubin; Baseline (Day -1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin; Day 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose; Baseline (Day -1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose; Day 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ketones; Baseline (Day -1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ketones; Day 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocyte esterase; Baseline (Day -1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocyte esterase; Day 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite; Baseline (Day -1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite; Day 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Occult blood; Baseline (Day -1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Occult blood; Day 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  pH; Baseline (Day -1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  pH; Day 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein; Baseline (Day -1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein; Day 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Specific gravity; Baseline (Day -1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Specific gravity; Day 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urobilinogen; Baseline (Day -1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urobilinogen; Day 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0

56. Primary Outcome: Part A: Number of Participants With Abnormal Findings for Urine Parameters in Cohort 2
Description: as for outcome 55
Time Frame: Baseline (Day -1) and Day 3
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 2 | 2 | 6 | 6
Participants
  Bilirubin; Baseline (Day -1) | 0 | 0 | 0 | 0
  Bilirubin; Day 3 | 0 | 0 | 0 | 0
  Glucose; Baseline (Day -1) | 0 | 0 | 0 | 0
  Glucose; Day 3 | 0 | 0 | 0 | 0
  Ketones; Baseline (Day -1) | 0 | 0 | 0 | 0
  Ketones; Day 3 | 0 | 0 | 0 | 0
  Leukocyte esterase; Baseline (Day -1) | 0 | 0 | 0 | 0
  Leukocyte esterase; Day 3 | 0 | 0 | 0 | 0
  Nitrite; Baseline (Day -1) | 0 | 0 | 0 | 0
  Nitrite; Day 3 | 0 | 0 | 0 | 0
  Occult blood; Baseline (Day -1) | 0 | 0 | 0 | 0
  Occult blood; Day 3 | 0 | 0 | 0 | 0
  pH; Baseline (Day -1) | 0 | 0 | 0 | 0
  pH; Day 3 | 0 | 0 | 0 | 0
  Protein; Baseline (Day -1) | 0 | 0 | 0 | 0
  Protein; Day 3 | 0 | 0 | 0 | 0
  Specific gravity; Baseline (Day -1) | 0 | 0 | 0 | 0
  Specific gravity; Day 3 | 0 | 0 | 0 | 0
  Urobilinogen; Baseline (Day -1) | 0 | 0 | 0 | 0
  Urobilinogen; Day 3 | 0 | 0 | 0 | 0

57. Primary Outcome: Part B: Number of Participants With Abnormal Findings for Urine Parameters
Description: Blood samples were collected for analysis of hematology parameters including Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, Leukocytes. Baseline is defined as the last available, non-missing assessment prior to the first administration of study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -2), Day 7, Day 15 and Follow-up (Day 25)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants
  Bilirubin; Baseline (Day -2) | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin; Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin; Day 15 | 0 | 0 | 0 | 0 | 0 | 2
  Bilirubin; Follow-up (Day 25) | 0 | 0 | 0 | 0 | 0 | 0
  Glucose; Baseline (Day -2) | 0 | 0 | 0 | 0 | 0 | 0
  Glucose; Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose; Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose; Follow-up (Day 25) | 0 | 0 | 0 | 0 | 0 | 0
  Ketones; Baseline (Day -2) | 1 | 2 | 0 | 0 | 0 | 0
  Ketones; Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Ketones; Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Ketones; Follow-up (Day 25) | 0 | 0 | 0 | 0 | 1 | 0
  Leukocyte esterase; Baseline (Day -2) | 0 | 0 | 0 | 0 | 0 | 1
  Leukocyte esterase; Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocyte esterase; Day 15 | 0 | 0 | 0 | 0 | 0 | 1
  Leukocyte esterase; Follow-up (Day 25) | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite; Baseline (Day -2) | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite; Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite; Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite; Follow-up (Day 25) | 0 | 0 | 0 | 0 | 0 | 0
  Occult blood; Baseline (Day -2) | 0 | 3 | 0 | 0 | 0 | 0
  Occult blood; Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Occult blood; Day 15 | 0 | 0 | 1 | 0 | 0 | 0
  Occult blood; Follow-up (Day 25) | 0 | 0 | 0 | 0 | 1 | 0
  pH; Baseline (Day -2) | 0 | 0 | 0 | 0 | 0 | 0
  pH; Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  pH; Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  pH; Follow-up (Day 25) | 0 | 0 | 0 | 0 | 0 | 0
  Protein; Baseline (Day -2) | 0 | 0 | 1 | 0 | 0 | 0
  Protein; Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Protein; Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Protein; Follow-up (Day 25) | 0 | 0 | 0 | 1 | 0 | 0
  Specific gravity; Baseline (Day -2) | 0 | 1 | 0 | 0 | 0 | 0
  Specific gravity; Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Specific gravity; Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Specific gravity; Follow-up (Day 25) | 0 | 0 | 0 | 0 | 0 | 0
  Urobilinogen; Baseline (Day -2) | 0 | 0 | 0 | 0 | 0 | 0
  Urobilinogen; Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Urobilinogen; Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Urobilinogen; Follow-up (Day 25) | 0 | 0 | 0 | 0 | 0 | 0

58. Primary Outcome: Part A: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Non-zero Concentration (AUC [0-t]) Following Single Dose Administration of GSK3352589
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-t) following administration of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part A was conducted by non-compartmental methods. The PK Parameter population comprised of all randomized participants who received at least one dose of active treatment and who had GSK3352589 Pharmacokinetic parameter estimates from any portion of the study.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36, 48 Hours Post-dose
Population: Pharmacokinetic Parameter Population comprised of all randomized participants who received at least one dose of active treatment and who had GSK3352589 Pharmacokinetic parameter estimates from any portion of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Nanogram per milliliter
Groups:
- Cohort 3: GSK3352589 150 mg: Participants received GSK3352589 150 mg tablet in Period 1 of Cohort 3 in Part A of the study.
- Cohort 3: GSK3352589 400 mg: Participants received GSK3352589 400 mg tablet in Period 2 of Cohort 3 in Part A of the study.
Arm/Group | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg | Cohort 3: GSK3352589 150 mg | Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 5
Hour*Nanogram per milliliter | 0.8452 (75.5) | 1.306 (66.2) | 2.480 (49.4) | 4.630 (63.9) | 2.771 (38.9) | 2.030 (24.4) | 9.416 (119.1) | 11.67 (124.7)

59. Primary Outcome: Part A: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC [0-infinity]) Following Single Dose Administration of GSK3352589
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-infinity) following administration of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part A was conducted by non-compartmental methods.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36, 48 Hours Post-dose
Population: Pharmacokinetic Parameter Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Nanogram per milliliter
Arm/Group | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg | Cohort 3: GSK3352589 150 mg | Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 3 | 5 | 6 | 2
Hour*Nanogram per milliliter | 0.9652 (83.7) | 1.446 (73.0) | 2.738 (46.3) | 5.031 (63.6) | 3.648 (53.3) | 2.372 (27.8) | 10.75 (119.1) | 17.49 (1.9)

60. Primary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) Following Single Dose Administration of GSK3352589
Description: Blood samples were collected from participants for pharmacokinetic analysis including Cmax following administration of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part A was conducted by non-compartmental methods.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36, 48 Hours Post-dose
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg | Cohort 3: GSK3352589 150 mg | Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 5
Nanogram per milliliter | 0.2339 (74.1) | 0.2919 (58.6) | 0.5541 (40.0) | 0.7318 (65.3) | 0.5397 (38.6) | 0.4317 (15.2) | 1.325 (111.6) | 1.157 (72.5)

61. Primary Outcome: Part A: Time to Reach Cmax (Tmax) Following Single Dose Administration of GSK3352589
Description: Blood samples were collected from participants for pharmacokinetic analysis including Tmax following administration of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part A was conducted by non-compartmental methods.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36, 48 Hours Post-dose
Population: Pharmacokinetic Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg | Cohort 3: GSK3352589 150 mg | Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 5
Hours | 1.25 [0.50 to 2.0] | 1.50 [1.0 to 3.0] | 1.00 [0.50 to 2.0] | 1.50 [1.0 to 4.0] | 1.25 [1.0 to 2.0] | 0.750 [0.50 to 2.0] | 1.25 [0.50 to 3.0] | 1.00 [0.50 to 4.0]

62. Primary Outcome: Part A: Terminal Elimination Half-life (t1/2) Following Single Dose Administration of GSK3352589
Description: Blood samples were collected from participants for pharmacokinetic analysis including t1/2 following administration of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part A was conducted by non-compartmental methods.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36, 48 Hours Post-dose
Population: Pharmacokinetic Parameter Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg | Cohort 3: GSK3352589 150 mg | Cohort 3: GSK3352589 400 mg
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 3 | 5 | 6 | 3
Hours | 5.54 (83.1) | 7.83 (65.1) | 17.1 (32.4) | 17.0 (11.8) | 19.2 (33.7) | 20.5 (19.7) | 16.1 (58.9) | 14.4 (39.7)

63. Primary Outcome: Part A: Cmax Following Single Dose Administration of GSK3352589-Food Effect
Description: Blood samples were collected from participants for pharmacokinetic analysis following administration of GSK3352589 in fasted and fed condition to assess the effect of food on pharmacokinetics of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part A was conducted by non-compartmental methods.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36, 48 Hours Post-dose
Population: Pharmacokinetic Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 6 | 6
Nanogram per milliliter | 0.5397 (38.6) | 0.4317 (15.2)
Statistical Analysis 1: Comparison: Part A: Cohort 2: GSK3352589 Fasted 25 mg vs Part A: Cohort 2: GSK3352589 Fed 25 mg; Test type: Other; p = 0.204, ANOVA; Ratio = 0.8000, 90% CI 2-sided [0.5940 to 1.077]

64. Primary Outcome: Part A: AUC (0-t) Following Single Dose Administration of GSK3352589- Food Effect
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-t) following administration of GSK3352589 in fasted and fed condition to assess the effect of food on pharmacokinetics of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part A was conducted by non-compartmental methods.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36, 48 Hours Post-dose
Population: Pharmacokinetic Parameter Population
Measure: Least Squares Mean (Standard Error); unit: Hours*Nanogram per milliliter
Arm/Group | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 6 | 6
Hours*Nanogram per milliliter | 1.019 (0.1287) | 0.7081 (0.1287)
Statistical Analysis 1: Comparison: Part A: Cohort 2: GSK3352589 Fasted 25 mg vs Part A: Cohort 2: GSK3352589 Fed 25 mg; Test type: Other; p = 0.118, ANOVA; Ratio = 0.7325, 90% CI 2-sided [0.5267 to 1.019]

65. Primary Outcome: Part A: AUC (0-infinity) Following Single Dose Administration of GSK3352589- Food Effect
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-infinity) following administration of GSK3352589 in fasted and fed condition to assess the effect of food on pharmacokinetics of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part A was conducted by non-compartmental methods.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36, 48 Hours Post-dose
Population: Pharmacokinetic Parameter Population
Measure: Least Squares Mean (Standard Error); unit: Hours*Nanogram per milliliter
Arm/Group | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 2: GSK3352589 Fed 25 mg
Number analyzed (Participants) | 6 | 6
Hours*Nanogram per milliliter | 1.294 (0.2105) | 0.8636 (0.1630)
Statistical Analysis 1: Comparison: Part A: Cohort 2: GSK3352589 Fasted 25 mg vs Part A: Cohort 2: GSK3352589 Fed 25 mg; Test type: Other; p = 0.157, ANOVA; Ratio = 0.6502, 90% CI 2-sided [0.3876 to 1.091]

66. Primary Outcome: Part B: AUC (0-t) Following Repeat Dose Administration of GSK3352589
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-t) following administration of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part B was conducted by non-compartmental methods.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 10, 11, 12, 14, 16, 24 Hours Post-dose on Day 1; Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 10, 11, 12, 14, 16, 24 Hours Post-dose on Day 14
Population: Pharmacokinetic Parameter Population. Only those participants with data available at specified time point were analyzed (reported by n=X in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Nanogram per milliliter
Arm/Group | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hour*Nanogram per milliliter
  Day 1; n=6, 6, 6, 6, 6 | 0.4479 (89.6) | 0.4647 (75.1) | 2.167 (41.2) | 3.459 (84.6) | 2.934 (90.0)
  Day 14; n=5, 6, 6, 6, 6: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Day 14; n=5, 6, 6, 6, 6 | 0.7147 (84.9) | 0.7176 (53.4) | 3.763 (21.5) | 6.121 (35.0) | 8.061 (53.9)

67. Primary Outcome: Part B: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to 24 Hours Post-dose (AUC [0-24]) Following Repeat Dose Administration of GSK3352589
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-24) following administration of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part B was conducted by non-compartmental methods.
Time Frame: as for outcome 66
Population: as for outcome 66
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Nanogram per milliliter
Arm/Group | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hour*Nanogram per milliliter
  Day 1; n=6, 6, 6, 6, 6 | 1.389 (58.6) | 1.641 (51.5) | 7.285 (40.6) | 11.41 (65.5) | 12.31 (73.3)
  Day 14; n=5, 6, 6, 6, 6: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Day 14; n=5, 6, 6, 6, 6 | 1.988 (62.5) | 1.970 (44.1) | 9.383 (23.2) | 15.73 (33.8) | 24.11 (45.9)

68. Primary Outcome: Part B: Area Under the Concentration-time Curve Over the Dosing Interval (AUC [0-tau]) Following Repeat Dose Administration of GSK3352589
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-tau) following administration of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part B was conducted by non-compartmental methods.
Time Frame: as for outcome 66
Population: as for outcome 66
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Nanogram per milliliter
Arm/Group | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hour*Nanogram per milliliter
  Day 1; n=6, 6, 6, 6, 6 | 0.5028 (87.9) | 0.5468 (72.9) | 2.522 (43.4) | 4.055 (80.0) | 3.673 (81.9)
  Day 14; n=5, 6, 6, 6, 6: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Day 14; n=5, 6, 6, 6, 6 | 0.8303 (82.7) | 0.8417 (53.8) | 4.421 (22.1) | 7.242 (34.9) | 9.914 (54.3)

69. Primary Outcome: Part B: Cmax Following Repeat Dose Administration of GSK3352589
Description: Blood samples were collected from participants for pharmacokinetic analysis including Cmax following administration of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part B was conducted by non-compartmental methods.
Time Frame: as for outcome 66
Population: as for outcome 66
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Nanogram per milliliter
  Day 1; n=6, 6, 6, 6, 6 | 0.1308 (93.0) | 0.1394 (51.2) | 0.5255 (17.9) | 0.8191 (78.5) | 0.6607 (67.4)
  Day 14; n=5, 6, 6, 6, 6: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Day 14; n=5, 6, 6, 6, 6 | 0.1655 (74.3) | 0.1919 (31.3) | 0.7149 (26.4) | 1.260 (36.7) | 1.526 (43.6)

70. Primary Outcome: Part B: Tmax Following Repeat Dose Administration of GSK3352589
Description: Blood samples were collected from participants for pharmacokinetic analysis including Tmax following administration of GSK3352589. Pharmacokinetic analysis of GSK3352589 in Part B was conducted by non-compartmental methods.
Time Frame: as for outcome 66
Population: as for outcome 66
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hours
  Day 1; n=6, 6, 6, 6, 6 | 0.767 [0.50 to 3.0] | 1.00 [0.50 to 3.0] | 1.00 [0.50 to 4.0] | 1.50 [0.50 to 3.0] | 0.750 [0.50 to 1.0]
  Day 14; n=5, 6, 6, 6, 6: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Day 14; n=5, 6, 6, 6, 6 | 0.500 [0.50 to 3.0] | 0.500 [0.50 to 3.0] | 1.50 [0.50 to 4.0] | 1.75 [0.50 to 2.5] | 0.500 [0.50 to 4.0]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-SAEs were collected up to 64 days in Cohort 1, up to 30 days in Cohort 2, up to 30 days in Cohort 3 each in Part A of the study and up to 25 days in Part B of the study.
Description: SAEs and non-SAEs were collected using Safety Population.
Groups:
- Part A: Cohort 1: Placebo: Participants received placebo tablet matching GSK3352589 orally in each Period of Cohort 1 in Part A of the study.
- Part A: Cohort 3: Placebo: Participants received placebo tablet matching GSK3352589 in each Period of Cohort 3 in Part A of the study.
Arm/Group | Part A: Cohort 1: Placebo | Part A: Cohort 1: GSK3352589 2 mg | Part A: Cohort 1: GSK3352589 5 mg | Part A: Cohort 1: GSK3352589 15 mg | Part A: Cohort 1: GSK3352589 50 mg | Part A: Cohort 2: Fasted Placebo | Part A: Cohort 2: Fed Placebo | Part A: Cohort 2: GSK3352589 Fed 25 mg | Part A: Cohort 2: GSK3352589 Fasted 25 mg | Part A: Cohort 3: Placebo | Part A: Cohort 3: GSK3352589 150 mg | Part A: Cohort 3: GSK3352589 400 mg | Part B: Placebo BID | Part B: GSK3352589 5 mg BID | Part B: GSK3352589 15 mg BID | Part B: GSK3352589 50 mg BID | Part B: GSK3352589 100 mg BID | Part B: GSK3352589 200 mg BID
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/5 | 0/2 | 0/2 | 0/6 | 0/6 | 0/4 | 0/6 | 0/5 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/6 | 0/6 | 0/6 | 0/5 | 0/2 | 0/2 | 0/6 | 0/6 | 0/4 | 0/6 | 0/5 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/8 | 5/6 | 3/6 | 2/6 | 2/5 | 1/2 | 0/2 | 3/6 | 1/6 | 2/4 | 3/6 | 1/5 | 9/10 | 5/6 | 6/6 | 2/6 | 5/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1: Placebo (N=8) | Part A: Cohort 1: GSK3352589 2 mg (N=6) | Part A: Cohort 1: GSK3352589 5 mg (N=6) | Part A: Cohort 1: GSK3352589 15 mg (N=6) | Part A: Cohort 1: GSK3352589 50 mg (N=5) | Part A: Cohort 2: Fasted Placebo (N=2) | Part A: Cohort 2: Fed Placebo (N=2) | Part A: Cohort 2: GSK3352589 Fed 25 mg (N=6) | Part A: Cohort 2: GSK3352589 Fasted 25 mg (N=6) | Part A: Cohort 3: Placebo (N=4) | Part A: Cohort 3: GSK3352589 150 mg (N=6) | Part A: Cohort 3: GSK3352589 400 mg (N=5) | Part B: Placebo BID (N=10) | Part B: GSK3352589 5 mg BID (N=6) | Part B: GSK3352589 15 mg BID (N=6) | Part B: GSK3352589 50 mg BID (N=6) | Part B: GSK3352589 100 mg BID (N=6) | Part B: GSK3352589 200 mg BID (N=6)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1: Placebo (N=8) | Part A: Cohort 1: GSK3352589 2 mg (N=6) | Part A: Cohort 1: GSK3352589 5 mg (N=6) | Part A: Cohort 1: GSK3352589 15 mg (N=6) | Part A: Cohort 1: GSK3352589 50 mg (N=5) | Part A: Cohort 2: Fasted Placebo (N=2) | Part A: Cohort 2: Fed Placebo (N=2) | Part A: Cohort 2: GSK3352589 Fed 25 mg (N=6) | Part A: Cohort 2: GSK3352589 Fasted 25 mg (N=6) | Part A: Cohort 3: Placebo (N=4) | Part A: Cohort 3: GSK3352589 150 mg (N=6) | Part A: Cohort 3: GSK3352589 400 mg (N=5) | Part B: Placebo BID (N=10) | Part B: GSK3352589 5 mg BID (N=6) | Part B: GSK3352589 15 mg BID (N=6) | Part B: GSK3352589 50 mg BID (N=6) | Part B: GSK3352589 100 mg BID (N=6) | Part B: GSK3352589 200 mg BID (N=6)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (6) | 2 (2) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hunger (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT03154086/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT03154086/SAP_001.pdf